CLINICAL TRIAL: NCT02918279
Title: Effect of Liraglutide for Weight Management in Pubertal Adolescent Subjects With Obesity. 56-week, Double-blind, Randomised, Parallel-group, Placebo-controlled Multi-national Trial Followed by a 26-week Period Off Study-drug
Brief Title: Effect of Liraglutide for Weight Management in Pubertal Adolescent Subjects With Obesity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN8022-4180; 2014-004353-14 (EudraCT Number); U1111-1162-7101 (Other: WHO)
Record Dates: First submitted 2016-09-27; First posted 2016-09-28 (Estimated); Results first posted 2020-04-27 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Metabolism and Nutrition Disorder; Obesity
MeSH Terms: conditions — Nutrition Disorders; Obesity | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liraglutide (Experimental)
  Interventions: Drug: Liraglutide
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Liraglutide — Administered once daily subcutaneously (s.c., under the skin)
  Arms: Liraglutide
Drug: Placebo — Administered once daily subcutaneously (s.c., under the skin)
  Arms: Placebo

SUMMARY:
This trial is conducted globally. The aim of this trial is to investigate the effect of liraglutide for weight management in pubertal adolescent subjects with obesity.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial
* Male or female, age 12 to less than 18 years at the time of signing informed consent and less than 18 years at date of randomisation
* BMI corresponding to equal to or above 30 kg/m^2 for adults by international cut-off points and equal or above the 95th percentile for age and sex (for diagnosis of obesity)
* Stable body weight during the previous 90 days before screening V2 (below 5 kg self-reported weight change)
* History of failing to lose sufficient weight with lifestyle modification as judged by the investigator and documented in subject's medical record

Exclusion Criteria:

* Pre-pubertal subjects (Tanner stage 1) at screening V2
* Type 1 diabetes mellitus (T1DM)
* Family or personal history of multiple endocrine neoplasia type 2 (MEN2)
* Medullary thyroid carcinoma (MTC)
* History of pancreatitis (acute or chronic)
* Subjects with secondary causes of obesity (i.e., hypothalamic, genetic or endocrine causes)
* Treatment with medications within 90 days before screening V2 that, based on the investigator's judgement, may cause significant weight change. This should also include treatment with any of the following medications: pramlintide, orlistat, zonisamide, topiramate, lorcaserin, phenteremine, bupropion, naltrexone, glucagon-like peptide-1 (GLP-1) receptor agonists, or metformin (used as treatment for obesity)
* Anti-diabetic treatment other than metformin
* History of major depressive disorder within 2 years before screening V2

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 251 (Actual)
Dates: Start 2016-09-29 (Actual); Primary Completion 2019-02-14 (Actual); Study Completion 2019-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR), Study Director — Novo Nordisk A/S
Locations (31):
- United States (12):
  - Novo Nordisk Investigational Site, Meridian, Idaho
  - Novo Nordisk Investigational Site, Baton Rouge, Louisiana
  - Novo Nordisk Investigational Site, Baltimore, Maryland
  - Novo Nordisk Investigational Site, Minneapolis, Minnesota
  - Novo Nordisk Investigational Site, Buffalo, New York
  - Novo Nordisk Investigational Site, Columbus, Ohio
  - Novo Nordisk Investigational Site, Dayton, Ohio
  - Novo Nordisk Investigational Site, Pittsburgh, Pennsylvania
  - Novo Nordisk Investigational Site, Charleston, South Carolina
  - Novo Nordisk Investigational Site, Goose Creek, South Carolina
  - Novo Nordisk Investigational Site, Greenville, South Carolina
  - Novo Nordisk Investigational Site, Memphis, Tennessee
- Belgium (5):
  - Novo Nordisk Investigational Site, Brussels
  - Novo Nordisk Investigational Site, Edegem
  - Novo Nordisk Investigational Site, Hasselt
  - Novo Nordisk Investigational Site, Leuven
  - Novo Nordisk Investigational Site, Namur
- Mexico (2):
  - Novo Nordisk Investigational Site, Ciudad Madero, Tamaulipas
  - Novo Nordisk Investigational Site, Puebla City
- Russia (8):
  - Novo Nordisk Investigational Site, Moscow
  - Novo Nordisk Investigational Site, Novosibirsk
  - Novo Nordisk Investigational Site, Rostov-on-Don
  - Novo Nordisk Investigational Site, Saint Petersburg
  - Novo Nordisk Investigational Site, Samara
  - Novo Nordisk Investigational Site, Stavropol
  - Novo Nordisk Investigational Site, Tomsk
  - Novo Nordisk Investigational Site, Ufa
- Sweden (4):
  - Novo Nordisk Investigational Site, Gothenburg
  - Novo Nordisk Investigational Site, Huddinge
  - Novo Nordisk Investigational Site, Malmo
  - Novo Nordisk Investigational Site, Uppsala

REFERENCES:
- [Result] Kelly AS, Auerbach P, Barrientos-Perez M, Gies I, Hale PM, Marcus C, Mastrandrea LD, Prabhu N, Arslanian S; NN8022-4180 Trial Investigators. A Randomized, Controlled Trial of Liraglutide for Adolescents with Obesity. N Engl J Med. 2020 May 28;382(22):2117-2128. doi: 10.1056/NEJMoa1916038. Epub 2020 Mar 31. PMID 32233338
- [Derived] Bensignor MO, Bramante CT, Bomberg EM, Fox CK, Hale PM, Kelly AS, Mamadi R, Prabhu N, Harder-Lauridsen NM, Gross AC. Evaluating potential predictors of weight loss response to liraglutide in adolescents with obesity: A post hoc analysis of the randomized, placebo-controlled SCALE Teens trial. Pediatr Obes. 2023 Sep;18(9):e13061. doi: 10.1111/ijpo.13061. Epub 2023 Jun 1. PMID 37264767

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted at 32 sites in 5 countries: Belgium (6 sites), Sweden (4 sites), Russia (8 sites), Mexico (2 sites) and the United States of America (USA - 12 sites). Additionally, 1 site in the USA was approved by the independent review board, but did not randomise any participant.
Pre-assignment Details: This trial consisted of a 12-week run-in period, during which participants received counselling on healthy nutrition and physical activity. Completed numbers include participants who completed the trial without prematurely discontinuing the trial product and participants who discontinued the trial product but came for the week 82 follow-up visit.
Groups:
- Liraglutide 3.0 mg: Participants received liraglutide in a dose escalation manner for 56 weeks: 0.6 mg during week 1, 1.2 mg during week 2, 1.8 mg during week 3, 2.4 mg during week 4 and 3.0 mg from week 5 to week 56. There was a 26-week off-study-drug follow-up period (week 57-82). Liraglutide was administered once daily by subcutaneous (s.c.; under the skin) injection in the abdomen, thigh or upper arm irrespective of the timing of meals.
- Placebo: Subjects received liraglutide matching placebo for 56 weeks. There was a 26-week off-study-drug follow-up period (week 57-82). Placebo for liraglutide was administered once daily by s.c. injection in the abdomen, thigh or upper arm irrespective of the timing of meals.
Period: Overall Study
Arm/Group | Liraglutide 3.0 mg | Placebo
Started | 125 | 126
Full Analysis Set | 125 | 126
Safety Analysis Set | 125 | 126
Completed | 112 | 103
Not Completed | 13 | 23
Not completed — Lost to Follow-up | 3 | 6
Not completed — Withdrawal by Subject | 5 | 15
Not completed — Withdrawal by parent/guardian | 2 | 1
Not completed — Other | 3 | 1

BASELINE CHARACTERISTICS:
Population: Results are based on the full analysis set (FAS) which included all randomised participants who had received at least one dose of trial product and had any post-randomisation data (according to the intention-to-treat [ITT] principle).
Groups:
- Liraglutide 3.0 mg: Participants received liraglutide in a dose escalation manner for 56 weeks: 0.6 mg during week 1, 1.2 mg during week 2, 1.8 mg during week 3, 2.4 mg during week 4 and 3.0 mg from week 5 to week 56. There was a 26-week off-study-drug follow-up period (week 57-82). Liraglutide was administered once daily by s.c. injection in the abdomen, thigh or upper arm irrespective of the timing of meals.
- Total: Total of all reporting groups
Arm/Group | Liraglutide 3.0 mg | Placebo | Total
Number analyzed (Participants) | 125 | 126 | 251
Age, Continuous [Mean (Standard Deviation); unit: Years] | 14.6 (1.6) | 14.5 (1.6) | 14.5 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 78 | 149
  Male | 54 | 48 | 102
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 32 | 24 | 56
  Not Hispanic or Latino | 93 | 102 | 195
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 0 | 2
  Black or African American | 14 | 6 | 20
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  White | 105 | 115 | 220
  Other | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change in BMI SDS (Week 0, Week 56)
Description: Change from baseline (week 0) in BMI SDS was evaluated at week 56. BMI SDS was calculated using the following formula: Z=[(value /M)^L - 1] / S*L; where L, M and S are median (M), skewness (L) and variation coefficient (S) of children/adolescents' BMI provided for each sex and age. For each subject, a standard deviation score Z (SDS) was calculated based on age and sex referring to the values L, M and S. The method is described in the world health organisation (WHO) Multicentre Growth Reference, which also contains the values for L, M and S by age and sex. For Z (SDS) scores below -3 and above 3, the score was adjusted as described in the WHO instruction. All available data were used for the analysis including data collected after treatment discontinuation. Results are based on both participants who completed the week 0-56 trial period and participants who prematurely discontinued the trial product but attended the follow-up visit at 56.
Time Frame: Week 0, week 56
Population: Results are based on the full analysis set (FAS) which included all randomised participants who had received at least one dose of trial product and had any post-randomisation data (according to the intention-to-treat [ITT] principle). "Overall Number of Participants Analyzed" = number of participants with available data.
Measure: Mean (Standard Deviation); unit: SDS score
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 113 | 105
SDS score | -0.25 (0.51) | -0.02 (0.54)
Statistical Analysis 1: Comparison: Liraglutide 3.0 mg vs Placebo; Analysis of in-trial data with missing observations was imputed from the placebo arm based on a jump to reference multiple (x100) imputation approach. Responses at week 56 were analysed using an analysis of covariance model with treatment, sex, region, baseline glycaemic category, stratification factor for Tanner stage and interaction between baseline glycaemic category and stratification factor for Tanner stage as fixed effects, baseline BMI SDS, age as covariates; Test type: Superiority; p = 0.0022, ANCOVA; Treatment difference = -0.22, 95% CI 2-sided [-0.37 to -0.08] — Liraglutide 3.0 mg - Placebo

2. Secondary Outcome: Percent of Subjects Achieving ≥5% Reduction in Baseline BMI
Description: Participants achieving more than or equal to 5% reduction in their baseline (week 0) BMI was evaluated at weeks 30, 56 and 82. Results are based on both participants who completed the trial period, week 0-30, week 0-56 or week 0-82, and participants who could not complete the corresponding trial period, but attended the follow-up visit at week 30, 56 or 82, respectively.
Time Frame: Weeks 30, 56 and 82
Population: Results are based on the FAS which included all randomised participants who had received at least one dose of trial product and had any post-randomisation data (according to the intention-to-treat [ITT] principle). "Overall Number of Participants Analyzed" = FAS. "Number Analyzed" = number of participants with available data.
Measure: Number; unit: Percentage of participants
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 125 | 126
Percentage of participants
  Week 30 (Yes): number analyzed (Participants) | 119 | 116
  Week 30 (Yes) | 46.2 | 14.7
  Week 30 (No): number analyzed (Participants) | 119 | 116
  Week 30 (No) | 53.8 | 85.3
  Week 56 (Yes): number analyzed (Participants) | 113 | 105
  Week 56 (Yes) | 45.1 | 19.0
  Week 56 (No): number analyzed (Participants) | 113 | 105
  Week 56 (No) | 54.9 | 81.0
  Week 82 (Yes): number analyzed (Participants) | 112 | 102
  Week 82 (Yes) | 29.5 | 18.6
  Week 82 (No): number analyzed (Participants) | 112 | 102
  Week 82 (No) | 70.5 | 81.4

3. Secondary Outcome: Percent of Subjects Achieving ≥10% Reduction in Baseline BMI
Description: Participants achieving more than or equal to 10% reduction in their baseline (week 0) BMI was evaluated at weeks 30, 56 and 82. Results are based on both participants who completed the trial period, week 0-30, week 0-56 or week 0-82, and participants who could not complete the corresponding trial period, but attended the follow-up visit at week 30, 56 or 82, respectively.
Time Frame: Weeks 30, 56 and 82
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 125 | 126
Percentage of participants
  Week 30 (Yes): number analyzed (Participants) | 119 | 116
  Week 30 (Yes) | 24.4 | 5.2
  Week 30 (No): number analyzed (Participants) | 119 | 116
  Week 30 (No) | 75.6 | 94.8
  Week 56 (Yes): number analyzed (Participants) | 113 | 105
  Week 56 (Yes) | 29.2 | 8.6
  Week 56 (No): number analyzed (Participants) | 113 | 105
  Week 56 (No) | 70.8 | 91.4
  Week 82 (Yes): number analyzed (Participants) | 112 | 102
  Week 82 (Yes) | 18.8 | 10.8
  Week 82 (No): number analyzed (Participants) | 112 | 102
  Week 82 (No) | 81.3 | 89.2

4. Secondary Outcome: Change in BMI SDS ((Week 0, Week 30); (Week 0, Week 82); (Week 56, Week 82))
Description: Change in BMI SDS was evaluated from baseline (week 0) to weeks 30 and 82, and from week 56 to week 82. BMI SDS was calculated using the following formula: Z=[(value /M)^L - 1] / S*L; where L, M and S are median (M), skewness (L) and variation coefficient (S) of children/adolescents' BMI provided for each sex and age. For each subject, a Z (SDS) score was calculated based on age and sex referring to the values L, M and S. The method is described in the WHO Multicentre Growth Reference, which also contains the values for L, M and S by age and sex. For Z (SDS) scores below -3 and above 3, the score was adjusted as described in the WHO instruction. All available data were used for the analysis including data collected after treatment discontinuation. Results are based on both participants who completed the trial period, week 0-30 or week 0-82, and participants who could not complete the corresponding trial period, but attended the follow-up visit at week 30 or 82, respectively.
Time Frame: (Week 0, week 30); (Week 0, week 82); (Week 56, week 82)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: SDS score
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 125 | 126
SDS score
  Change from week 0 to week 30: number analyzed (Participants) | 119 | 116
  Change from week 0 to week 30 | -0.26 (0.34) | -0.04 (0.33)
  Change from week 0 to week 82: number analyzed (Participants) | 112 | 102
  Change from week 0 to week 82 | -0.06 (0.53) | 0.07 (0.66)
  Change from week 56 to week 82: number analyzed (Participants) | 99 | 98
  Change from week 56 to week 82 | 0.22 (0.28) | 0.08 (0.27)

5. Secondary Outcome: Change in BMI
Description: Change in BMI was evaluated from baseline (week 0) to weeks 30 and 56, and from week 56 to week 82. Results are based on both participants who completed the trial period, week 0-30, week 0-56 or week 0-82, and participants who could not complete the corresponding trial period, but attended the follow-up visit at week 30, 56 or 82, respectively.
Time Frame: (Week 0, week 30); (Week 0, week 56); (Week 56, week 82)
Population: Results are based on the FAS which included all randomised participants who had received at least one dose of trial product and had any post-randomisation data (according to the ITT principle). "Overall Number of Participants Analyzed" = FAS. "Number Analyzed" = number of participants with available data.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 125 | 126
kg/m^2
  Change from week 0 to week 30: number analyzed (Participants) | 119 | 116
  Change from week 0 to week 30 | -1.8 (2.1) | -0.2 (2.2)
  Change from week 0 to week 56: number analyzed (Participants) | 113 | 105
  Change from week 0 to week 56 | -1.6 (3.1) | 0.1 (3.4)
  Change from week 56 to week 82: number analyzed (Participants) | 99 | 98
  Change from week 56 to week 82 | 1.5 (1.7) | 0.7 (1.7)

6. Secondary Outcome: Change in Body Weight (kg)
Description: Change in body weight (kg) was evaluated from baseline (week 0) to weeks 30 and 56, and from week 56 to week 82. Results are based on both participants who completed the trial period, week 0-30, week 0-56 or week 0-82, and participants who could not complete the corresponding trial period, but attended the follow-up visit at week 30, 56 or 82, respectively.
Time Frame: (Week 0, week 30); (Week 0, week 56); (Week 56, week 82)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 125 | 126
kg
  Change from week 0 to week 30: number analyzed (Participants) | 119 | 116
  Change from week 0 to week 30 | -3.9 (6.1) | 0.4 (6.6)
  Change from week 0 to week 56: number analyzed (Participants) | 113 | 105
  Change from week 0 to week 56 | -2.7 (9.1) | 2.1 (10.2)
  Change from week 56 to week 82: number analyzed (Participants) | 99 | 98
  Change from week 56 to week 82 | 4.7 (4.6) | 2.4 (4.9)

7. Secondary Outcome: Change in Body Weight (%)
Description: Relative change in body weight (kg) was evaluated from baseline (week 0) to weeks 30 and 56, and from week 56 to week 82. Results are based on both participants who completed the trial period, week 0-30, week 0-56 or week 0-82, and participants who could not complete the corresponding trial period, but attended the follow-up visit at week 30, 56 or 82, respectively.
Time Frame: (Week 0, week 30); (Week 0, week 56); (Week 56, week 82)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 125 | 126
Percentage change
  Change from week 0 to week 30: number analyzed (Participants) | 119 | 116
  Change from week 0 to week 30 | -4.3 (6.5) | 0.4 (6.2)
  Change from week 0 to week 56: number analyzed (Participants) | 113 | 105
  Change from week 0 to week 56 | -3.2 (9.4) | 2.2 (9.5)
  Change from week 56 to week 82: number analyzed (Participants) | 99 | 98
  Change from week 56 to week 82 | 5.3 (5.7) | 2.3 (4.9)

8. Secondary Outcome: Change in Body Weight (lb)
Description: Body weight was not analysed in pounds (lb). It was analysed for standard unit, 'kg' only.
Time Frame: (Week 0, week 30); (Week 0, week 56); (Week 56, week 82)
Population: Body weight was not analysed in pounds (lb).
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Change in Waist Circumference
Description: Change in waist circumference was evaluated from baseline (week 0) to weeks 30 and 56, and from week 56 to week 82. Results are based on the participants who completed the corresponding trial period, week 0-30, week 0-56 or week 0-82.
Time Frame: (Week 0, week 30); (Week 0, week 56); (Week 56, week 82)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 125 | 126
cm
  Change from week 0 to week 30: number analyzed (Participants) | 116 | 114
  Change from week 0 to week 30 | -4.63 (6.24) | -2.01 (5.94)
  Change from week 0 to week 56: number analyzed (Participants) | 100 | 101
  Change from week 0 to week 56 | -5.12 (7.87) | -1.51 (8.20)
  Change from week 56 to week 82: number analyzed (Participants) | 98 | 98
  Change from week 56 to week 82 | 3.58 (4.30) | 1.24 (5.60)

10. Secondary Outcome: Change in Waist-to-hip Circumference Ratio
Description: Change in waist-to-hip circumference ratio was evaluated from baseline (week 0) to weeks 30 and 56, and from week 56 to week 82. Results are based on the participants who completed the corresponding trial period, week 0-30, week 0-56 or week 0-82.
Time Frame: (Week 0, week 30); (Week 0, week 56); (Week 56, week 82)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 125 | 126
Ratio
  Change from week 0 to week 30: number analyzed (Participants) | 116 | 114
  Change from week 0 to week 30 | -0.015 (0.042) | -0.018 (0.042)
  Change from week 0 to week 56: number analyzed (Participants) | 100 | 100
  Change from week 0 to week 56 | -0.022 (0.053) | -0.023 (0.051)
  Change from week 56 to week 82: number analyzed (Participants) | 98 | 97
  Change from week 56 to week 82 | 0.010 (0.031) | 0.003 (0.049)

11. Secondary Outcome: Change in hsCRP
Description: Change in high sensitivity C reactive protein (hsCRP) was evaluated from baseline (week 0) to weeks 30 and 56, and from week 56 to week 82. Results are based on the participants who completed the corresponding trial period, week 0-30, week 0-56 or week 0-82.
Time Frame: (Week 0, week 30); (Week 0, week 56); (Week 56, week 82)
Population: Results are based on the safety analysis set (SAS) which included all randomised participants exposed to at least one dose of trial product. "Overall Number of Participants Analyzed" = SAS. "Number Analyzed" = number of participants with available data.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 125 | 126
mg/L
  Change from week 0 to week 30: number analyzed (Participants) | 116 | 116
  Change from week 0 to week 30 | -0.22 (5.04) | -0.56 (4.68)
  Change from week 0 to week 56: number analyzed (Participants) | 105 | 101
  Change from week 0 to week 56 | -0.25 (4.54) | -0.14 (3.44)
  Change from week 56 to week 82: number analyzed (Participants) | 99 | 97
  Change from week 56 to week 82 | 1.51 (7.61) | 1.00 (4.22)

12. Secondary Outcome: Change in Fasting Lipid: Total Cholesterol (Ratio to Baseline)
Description: Change in total cholesterol from baseline (week 0) to weeks 30 and 56, and from week 56 to week 82 are presented as ratio to baseline. Results are based on the participants who completed the corresponding trial period, week 0-30, week 0-56 or week 0-82.
Time Frame: (Week 0, week 30); (Week 0, week 56); (Week 56, week 82)
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of total cholesterol
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 125 | 126
Ratio of total cholesterol
  Change from week 0 to week 30: number analyzed (Participants) | 116 | 116
  Change from week 0 to week 30 | 1.00 (12.8) | 0.98 (13.0)
  Change from week 0 to week 56: number analyzed (Participants) | 105 | 101
  Change from week 0 to week 56 | 1.00 (14.2) | 1.00 (13.0)
  Change from week 56 to week 82: number analyzed (Participants) | 99 | 97
  Change from week 56 to week 82 | 1.02 (14.7) | 1.02 (14.9)

13. Secondary Outcome: Change in Fasting Lipid: LDL-cholesterol (Ratio to Baseline)
Description: Change in low density lipoprotein (LDL) cholesterol from baseline (week 0) to weeks 30 and 56, and from week 56 to week 82 are presented as ratio to baseline. Results are based on the participants who completed the corresponding trial period, week 0-30, week 0-56 or week 0-82.
Time Frame: (Week 0, week 30); (Week 0, week 56); (Week 56, week 82)
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of LDL-cholesterol
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 125 | 126
Ratio of LDL-cholesterol
  Change from week 0 to week 30: number analyzed (Participants) | 116 | 116
  Change from week 0 to week 30 | 1.00 (19.8) | 1.00 (26.1)
  Change from week 0 to week 56: number analyzed (Participants) | 105 | 101
  Change from week 0 to week 56 | 0.99 (21.8) | 1.02 (23.6)
  Change from week 56 to week 82: number analyzed (Participants) | 99 | 97
  Change from week 56 to week 82 | 1.03 (22.5) | 1.04 (20.6)

14. Secondary Outcome: Change in Fasting Lipid: HDL-cholesterol (Ratio to Baseline)
Description: Change in high density lipoprotein (HDL) cholesterol from baseline (week 0) to weeks 30 and 56, and from week 56 to week 82 are presented as ratio to baseline. Results are based on the participants who completed the corresponding trial period, week 0-30, week 0-56 or week 0-82.
Time Frame: (Week 0, week 30); (Week 0, week 56); (Week 56, week 82)
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of HDL-cholesterol
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 125 | 126
Ratio of HDL-cholesterol
  Change from week 0 to week 30: number analyzed (Participants) | 116 | 116
  Change from week 0 to week 30 | 1.04 (15.3) | 1.01 (20.5)
  Change from week 0 to week 56: number analyzed (Participants) | 105 | 101
  Change from week 0 to week 56 | 1.04 (17.4) | 1.02 (18.9)
  Change from week 56 to week 82: number analyzed (Participants) | 99 | 97
  Change from week 56 to week 82 | 0.99 (15.8) | 1.00 (15.2)

15. Secondary Outcome: Change in Fasting Lipid: Non-HDL Cholesterol (Ratio to Baseline)
Description: Change in non-HDL cholesterol from baseline (week 0) to weeks 30 and 56, and from week 56 to week 82 are presented as ratio to baseline. Results are based on the participants who completed the corresponding trial period, week 0-30, week 0-56 or week 0-82.
Time Frame: (Week 0, week 30); (Week 0, week 56); (Week 56, week 82)
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of non-HDL cholesterol
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 125 | 126
Ratio of non-HDL cholesterol
  Change from week 0 to week 30: number analyzed (Participants) | 116 | 116
  Change from week 0 to week 30 | 0.98 (16.8) | 0.97 (18.0)
  Change from week 0 to week 56: number analyzed (Participants) | 105 | 101
  Change from week 0 to week 56 | 0.98 (18.4) | 0.99 (16.7)
  Change from week 56 to week 82: number analyzed (Participants) | 99 | 97
  Change from week 56 to week 82 | 1.03 (19.8) | 1.02 (18.6)

16. Secondary Outcome: Change in Fasting Lipid: VLDL Cholesterol (Ratio to Baseline)
Description: Change in very low density lipoprotein (VLDL) cholesterol from baseline (week 0) to weeks 30 and 56, and from week 56 to week 82 are presented as ratio to baseline. Results are based on the participants who completed the corresponding trial period, week 0-30, week 0-56 or week 0-82.
Time Frame: (Week 0, week 30); (Week 0, week 56); (Week 56, week 82)
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of VLDL cholesterol
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 125 | 126
Ratio of VLDL cholesterol
  Change from week 0 to week 30: number analyzed (Participants) | 116 | 116
  Change from week 0 to week 30 | 0.91 (36.8) | 0.90 (42.7)
  Change from week 0 to week 56: number analyzed (Participants) | 105 | 101
  Change from week 0 to week 56 | 0.92 (43.7) | 0.93 (34.6)
  Change from week 56 to week 82: number analyzed (Participants) | 99 | 97
  Change from week 56 to week 82 | 1.04 (51.0) | 0.97 (34.1)

17. Secondary Outcome: Change in Fasting Lipid: Triglycerides (Ratio to Baseline)
Description: Change in triglycerides from baseline (week 0) to weeks 30 and 56, and from week 56 to week 82 are presented as ratio to baseline. Results are based on the participants who completed the corresponding trial period, week 0-30, week 0-56 or week 0-82.
Time Frame: (Week 0, week 30); (Week 0, week 56); (Week 56, week 82)
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of triglycerides
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 125 | 126
Ratio of triglycerides
  Change from week 0 to week 30: number analyzed (Participants) | 116 | 116
  Change from week 0 to week 30 | 0.91 (36.9) | 0.91 (42.9)
  Change from week 0 to week 56: number analyzed (Participants) | 105 | 101
  Change from week 0 to week 56 | 0.92 (43.2) | 0.93 (34.4)
  Change from week 56 to week 82: number analyzed (Participants) | 99 | 97
  Change from week 56 to week 82 | 1.04 (50.4) | 0.97 (34.0)

18. Secondary Outcome: Change in Fasting Lipid: FFA (Ratio to Baseline)
Description: Change in free fatty acids (FFA) from baseline (week 0) to weeks 30 and 56, and from week 56 to week 82 are presented as ratio to baseline. Results are based on the participants who completed the corresponding trial period, week 0-30, week 0-56 or week 0-82.
Time Frame: (Week 0, week 30); (Week 0, week 56); (Week 56, week 82)
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of FFA
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 125 | 126
Ratio of FFA
  Change from week 0 to week 30: number analyzed (Participants) | 116 | 113
  Change from week 0 to week 30 | 0.96 (57.7) | 0.83 (56.4)
  Change from week 0 to week 56: number analyzed (Participants) | 105 | 100
  Change from week 0 to week 56 | 1.00 (48.9) | 0.95 (50.8)
  Change from week 56 to week 82: number analyzed (Participants) | 99 | 97
  Change from week 56 to week 82 | 0.99 (55.2) | 0.94 (38.0)

19. Secondary Outcome: Change in Systolic and Diastolic Blood Pressure
Description: Change in systolic blood pressure (SBP) and diastolic blood pressure (DBP) was evaluated from baseline (week 0) to weeks 30 and 56, and from week 56 to week 82. Results are based on the participants who completed the corresponding trial period, week 0-30, week 0-56 or week 0-82.
Time Frame: (Week 0, week 30); (Week 0, week 56); (Week 56, week 82)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 125 | 126
mmHg
  SBP: Change from week 0 to week 30: number analyzed (Participants) | 116 | 114
  SBP: Change from week 0 to week 30 | -2 (9) | -1 (10)
  SBP: Change from week 0 to week 56: number analyzed (Participants) | 102 | 101
  SBP: Change from week 0 to week 56 | -2 (10) | 1 (10)
  SBP: Change from week 56 to week 82: number analyzed (Participants) | 99 | 98
  SBP: Change from week 56 to week 82 | 2 (9) | 1 (10)
  DBP: Change from week 0 to week 30: number analyzed (Participants) | 116 | 114
  DBP: Change from week 0 to week 30 | -0 (8) | -1 (10)
  DBP: Change from week 0 to week 56: number analyzed (Participants) | 102 | 101
  DBP: Change from week 0 to week 56 | 1 (9) | -1 (9)
  DBP: Change from week 56 to week 82: number analyzed (Participants) | 99 | 98
  DBP: Change from week 56 to week 82 | 2 (8) | 2 (7)

20. Secondary Outcome: Change in HbA1c
Description: Change in glycosylated haemoglobin (HbA1c) was evaluated from baseline (week 0) to weeks 30 and 56, and from week 56 to week 82. Results are based on the participants who completed the corresponding trial period, week 0-30, week 0-56 or week 0-82.
Time Frame: (Week 0, week 30); (Week 0, week 56); (Week 56, week 82)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 125 | 126
Percentage of HbA1c
  Change from week 0 to week 30: number analyzed (Participants) | 115 | 116
  Change from week 0 to week 30 | -0.1 (0.3) | -0.0 (0.3)
  Change from week 0 to week 56: number analyzed (Participants) | 105 | 101
  Change from week 0 to week 56 | -0.1 (0.3) | -0.0 (0.2)
  Change from week 56 to week 82: number analyzed (Participants) | 99 | 97
  Change from week 56 to week 82 | 0.1 (0.2) | 0.1 (0.3)

21. Secondary Outcome: Change in FPG
Description: Change in fasting plasma glucose (FPG) was evaluated from baseline (week 0) to weeks 30 and 56, and from week 56 to week 82. Results are based on the participants who completed treatment for the corresponding treatment period (week 0-30, week 0-56 or week 0-82).
Time Frame: (Week 0, week 30); (Week 0, week 56); (Week 56, week 82)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 125 | 126
mmol/L
  Change from week 0 to week 30: number analyzed (Participants) | 116 | 114
  Change from week 0 to week 30 | -0.2 (0.4) | -0.0 (0.5)
  Change from week 0 to week 56: number analyzed (Participants) | 105 | 100
  Change from week 0 to week 56 | -0.1 (0.5) | -0.0 (0.6)
  Change from week 56 to week 82: number analyzed (Participants) | 99 | 95
  Change from week 56 to week 82 | 0.1 (0.6) | 0.1 (0.5)

22. Secondary Outcome: Change in Fasting Insulin (Ratio to Baseline)
Description: Change in fasting insulin from baseline (week 0) to weeks 30 and 56, and from week 56 to week 82 are presented as ratio to baseline. Results are based on the participants who completed the corresponding trial period, week 0-30, week 0-56 or week 0-82.
Time Frame: (Week 0, week 30); (Week 0, week 56); (Week 56, week 82)
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of fasting insulin
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 125 | 126
Ratio of fasting insulin
  Change from week 0 to week 30: number analyzed (Participants) | 114 | 112
  Change from week 0 to week 30 | 1.13 (70.9) | 1.14 (53.7)
  Change from week 0 to week 56: number analyzed (Participants) | 105 | 101
  Change from week 0 to week 56 | 1.06 (69.4) | 1.10 (73.8)
  Change from week 56 to week 82: number analyzed (Participants) | 98 | 97
  Change from week 56 to week 82 | 1.00 (60.9) | 1.08 (55.2)

23. Secondary Outcome: Change in Fasting C-peptide (Ratio to Baseline)
Description: Change in fasting C-peptide from baseline (week 0) to weeks 30 and 56, and from week 56 to week 82 are presented as ratio to baseline. Results are based on the participants who completed the corresponding trial period, week 0-30, week 0-56 or week 0-82.
Time Frame: (Week 0, week 30); (Week 0, week 56); (Week 56, week 82)
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of fasting C-peptide
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 125 | 126
Ratio of fasting C-peptide
  Change from week 0 to week 30: number analyzed (Participants) | 114 | 112
  Change from week 0 to week 30 | 1.12 (42.6) | 1.04 (35.1)
  Change from week 0 to week 56: number analyzed (Participants) | 105 | 100
  Change from week 0 to week 56 | 0.98 (44.9) | 0.97 (47.4)
  Change from week 56 to week 82: number analyzed (Participants) | 98 | 96
  Change from week 56 to week 82 | 0.92 (43.6) | 0.94 (32.9)

24. Secondary Outcome: Change in Glycaemic Category
Description: Number of participants in glycaemic categories, "normoglycaemia, pre-diabetes and type 2 diabetes (T2DM)" at baseline (weeks -2), and weeks 30, 56 and 82 are presented. These categories were set as per the following criteria: 1) Normoglycaemia: FPG <5.6 mmol/L (<100 mg/dL) and/or HbA1c <5.7%. 2) Pre-diabetes: FPG 5.6-6.9 mmol/L (both inclusive), FPG 100-125 mg/dL (both inclusive) or HbA1c 5.7-6.4% (both inclusive). 3) Type 2 diabetes (T2DM): FPG ≥7.0 mmol/L (≥126 mg/dL) and/or HbA1c ≥6.5%. Week 30, 56 and 82 results are based on the participants who completed the corresponding trial period, week 0-30, week 0-56 or week 0-82.
Time Frame: Week -2, week 30, week 56 and week 82
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 125 | 126
Participants
  Week -2: Normoglycaemia | 93 | 93
  Week -2: Pre-diabetes | 31 | 32
  Week -2: Type 2 diabetes | 1 | 1
  Week 30: number analyzed (Participants) | 116 | 116
  Week 30: Normoglycaemia | 95 | 86
  Week 30: Pre-diabetes | 19 | 29
  Week 30: Type 2 diabetes | 2 | 1
  Week 56: number analyzed (Participants) | 105 | 101
  Week 56: Normoglycaemia | 86 | 75
  Week 56: Pre-diabetes | 17 | 24
  Week 56: Type 2 diabetes | 2 | 2
  Week 82: number analyzed (Participants) | 100 | 99
  Week 82: Normoglycaemia | 79 | 65
  Week 82: Pre-diabetes | 20 | 30
  Week 82: Type 2 diabetes | 1 | 4

25. Secondary Outcome: Change in HOMA-B (Ratio to Baseline)
Description: Change in homeostasis model assessment of beta-cell function (HOMA-B) from baseline (week 0) to weeks 30 and 56, and from week 56 to week 82 are presented as ratio to baseline. HOMA-B was calculated as: Beta-cell function (%) = 20·fasting insulin[mU/L]/(FPG[mmol/L]-3.5). Results are based on the participants who completed the corresponding trial period, week 0-30, week 0-56 or week 0-82.
Time Frame: (Week 0, week 30); (Week 0, week 56); (Week 56, week 82)
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of HOMA-B
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 125 | 126
Ratio of HOMA-B
  Change from week 0 to week 30: number analyzed (Participants) | 114 | 110
  Change from week 0 to week 30 | 1.32 (70.8) | 1.17 (59.5)
  Change from week 0 to week 56: number analyzed (Participants) | 105 | 100
  Change from week 0 to week 56 | 1.13 (67.0) | 1.11 (58.0)
  Change from week 56 to week 82: number analyzed (Participants) | 98 | 95
  Change from week 56 to week 82 | 0.92 (65.9) | 1.02 (50.2)

26. Secondary Outcome: Change in HOMA-IR (Ratio to Baseline)
Description: Change in homeostasis model assessment of insulin resistance (HOMA-IR) from baseline (week 0) to weeks 30 and 56, and from week 56 to week 82 are presented as ratio to baseline. HOMA-IR was calculated as: Insulin resistance (%) = fasting insulin [mU/L] x FPG [mmol/L]/ 22.5. Results are based on the participants who completed the corresponding trial period, week 0-30, week 0-56 or week 0-82.
Time Frame: (Week 0, week 30); (Week 0, week 56); (Week 56, week 82)
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of HOMA-IR
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 125 | 126
Ratio of HOMA-IR
  Change from week 0 to week 30: number analyzed (Participants) | 114 | 110
  Change from week 0 to week 30 | 1.08 (75.2) | 1.14 (55.6)
  Change from week 0 to week 56: number analyzed (Participants) | 105 | 100
  Change from week 0 to week 56 | 1.04 (75.3) | 1.09 (80.0)
  Change from week 56 to week 82: number analyzed (Participants) | 98 | 95
  Change from week 56 to week 82 | 1.03 (64.2) | 1.11 (60.5)

27. Secondary Outcome: Change in IWQOL-Kids
Description: Change in Impact of Weight on Quality of Life-Kids (IWQOL-Kids) was evaluated from baseline (week 0) to weeks 30 and 56, and from week 56 to week 82. The IWQOL-Kids is a 27-item measure of weight-related quality of life. There are four domain scores (Physical Comfort, Body Esteem, Social Life and Family Life) and a total score. Scores for all domains and total score range from 0-100, with higher scores representing better health-related quality of life. IWQOL-kids data at week 82 was not collected, thus could not be evaluated. Results are based on the participants who completed the corresponding trial period, week 0-30, week 0-56 or week 0-82.
Time Frame: (Week 0, week 30); (Week 0, week 56); (Week 56, week 82)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 125 | 126
Scores on a scale
  Body Esteem: Change from week 0 to week 30: number analyzed (Participants) | 112 | 116
  Body Esteem: Change from week 0 to week 30 | 10.62 (19.88) | 6.73 (26.87)
  Body Esteem: Change from week 0 to week 56: number analyzed (Participants) | 104 | 99
  Body Esteem: Change from week 0 to week 56 | 13.33 (19.47) | 13.24 (22.72)
  Body Esteem: Change from week 56 to week 82: number analyzed (Participants) | 0 | 0
  Family Relation: Change from week 0 to week 30: number analyzed (Participants) | 112 | 116
  Family Relation: Change from week 0 to week 30 | 2.53 (9.66) | -2.19 (17.53)
  Family Relation: Change from week 0 to week 56: number analyzed (Participants) | 104 | 99
  Family Relation: Change from week 0 to week 56 | 1.44 (14.31) | 0.97 (5.61)
  Family Relation: Change from week 56 to week 82: number analyzed (Participants) | 0 | 0
  Physical Function: Change from week 0 to week 30: number analyzed (Participants) | 112 | 116
  Physical Function: Change from week 0 to week 30 | 3.94 (15.34) | 0.43 (22.02)
  Physical Function: Change from week 0 to week 56: number analyzed (Participants) | 104 | 99
  Physical Function: Change from week 0 to week 56 | 6.17 (15.44) | 3.32 (16.60)
  Physical Function: Change from week 56 to week 82: number analyzed (Participants) | 0 | 0
  Social Life: Change from week 0 to week 30: number analyzed (Participants) | 112 | 116
  Social Life: Change from week 0 to week 30 | 5.32 (10.56) | 1.76 (21.98)
  Social Life: Change from week 0 to week 56: number analyzed (Participants) | 104 | 99
  Social Life: Change from week 0 to week 56 | 5.97 (19.48) | 6.06 (14.04)
  Social Life: Change from week 56 to week 82: number analyzed (Participants) | 0 | 0
  Total: Change from week 0 to week 30: number analyzed (Participants) | 112 | 116
  Total: Change from week 0 to week 30 | 6.16 (11.04) | 2.24 (19.69)
  Total: Change from week 0 to week 56: number analyzed (Participants) | 104 | 99
  Total: Change from week 0 to week 56 | 7.46 (13.70) | 6.72 (11.62)
  Total: Change from week 56 to week 82: number analyzed (Participants) | 0 | 0

28. Secondary Outcome: Change in BMI SDS (%)
Description: Relative change in BMI SDS was evaluated from baseline (week 0) to weeks 30 and 56. Results are based on the participants who completed the corresponding trial period, week 0-30 or week 0-56.
Time Frame: (Week 0, week 30); (Week 0, week 56)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percentage change
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 125 | 126
Percentage change
  Change from week 0 to week 30: number analyzed (Participants) | 119 | 116
  Change from week 0 to week 30 | -8.73 (1.05) | -1.70 (1.07)
  Change from week 0 to week 56: number analyzed (Participants) | 113 | 105
  Change from week 0 to week 56 | -8.32 (1.68) | -0.68 (1.74)

29. Secondary Outcome: Change in Nutritional Compliance
Description: This outcome measure presents "nutritional compliance results" recorded at baseline (week 0), week 30 and week 56. Nutritional compliance was recorded on a 0 to 10 numeric rating scale, with higher scores representing better compliance. Week 30 and 56 results are based on the participants who completed the corresponding trial period, week 0-30 or week 0-56.
Time Frame: Week 0, week 30 and week 56
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 125 | 126
Score on a scale
  Week 0: number analyzed (Participants) | 123 | 126
  Week 0 | 7.10 (1.74) | 7.07 (1.69)
  Week 30: number analyzed (Participants) | 114 | 114
  Week 30 | 6.74 (2.08) | 6.51 (1.91)
  Week 56: number analyzed (Participants) | 100 | 101
  Week 56 | 6.87 (1.87) | 6.45 (1.84)

30. Secondary Outcome: Number of Treatment Emergent Adverse Events
Description: A treatment emergent adverse event (TEAE) was defined as an event that occurred in the "on-treatment" period. 'On-treatment' period: Events with onset date between the first day of trial product administration and any of the following date, whichever came first: 1) 14 days after the last day on trial product, or 2) follow-up visit (week 58) for participants who discontinued trial product, or 3) last study visit (participants withdrawn without follow-up visit).
Time Frame: Week 0-56 + 14 days
Population: Results are based on the SAS which included all randomised participants exposed to at least one dose of trial product. "Overall Number of Participants Analyzed" = SAS.
Measure: Number; unit: Events
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 125 | 126
Events | 777 | 627

31. Secondary Outcome: Number of Treatment Emergent Hypoglycaemic Episodes (ADA/ISPAD Classification)
Description: A hypoglycaemic episode was defined as treatment emergent if the onset of the episode was on or after the first day of exposure to randomised treatment and no later than 14 days after the last day on randomised treatment. Severe hypoglycaemia episodes were recorded as per international society for pediatric and adolescent diabetes (ISPAD) definition. And the following presented hypoglycaemia episodes were recorded as per American Diabetes Association (ADA) definition: asymptomatic hypoglycaemia, documented symptomatic hypoglycaemia, pseudo-hypoglycaemia and probable symptomatic hypoglycaemia.
Time Frame: Week 0-56 + 14 days
Population: as for outcome 30
Measure: Number; unit: Episodes
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 125 | 126
Episodes
  Severe hypoglycaemia | 0 | 0
  Asymptomatic hypoglycaemia | 12 | 17
  Documented symptomatic hypoglycaemia | 31 | 6
  Probable symptomatic hypoglycaemia | 1 | 2
  Pseudo-hypoglycaemia | 30 | 3
  Unclassifiable | 4 | 0

32. Secondary Outcome: Number of Treatment Emergent Hypoglycaemic Episodes (Novo Nordisk/ISPAD Classification)
Description: Severe hypoglycaemia episodes were recorded as per the ISPAD definition. And the following presented hypoglycaemia episodes were recorded as per Novo Nordisk definition: Symptomatic BG-confirmed: An episode that is blood glucose (BG) confirmed by plasma glucose (PG) value <3.1 mmol/L with symptoms consistent with hypoglycaemia. Asymptomatic BG-confirmed: An episode that is BG-confirmed by PG value <3.1 mmol/L without symptoms consistent with hypoglycaemia. 4) Severe or BG-confirmed symptomatic: An episode that is severe according to the ISPAD classification or BG-confirmed by a PG value <3.1 mmol/L with symptoms consistent with hypoglycaemia. 5) BG-confirmed: An episode that is BG-confirmed by a PG value <3.1 mmol/L with or without symptoms consistent with hypoglycaemia. 6) Severe or BG-confirmed: An episode that is severe according to the ISPAD classification or BG-confirmed by a PG value <3.1 mmol/L with or without symptoms consistent with hypoglycaemia.
Time Frame: Week 0-56 + 14 days
Population: as for outcome 30
Measure: Number; unit: Episodes
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 125 | 126
Episodes
  Severe hypoglycaemia | 0 | 0
  Asymptomatic BG-confirmed hypoglycaemia | 1 | 1
  Symptomatic BG-confirmed hypoglycaemia | 4 | 0
  Unclassifiable | 73 | 27

33. Secondary Outcome: Occurrence of Anti-liraglutide Antibodies
Description: This outcome measure is only applicable for the liraglutide 3.0 mg treatment arm. Number of participants who measured with anti-liraglutide binding antibodies at weeks 0, 30, 56, 58, 70 and 82 are presented.
Time Frame: Weeks 0, 30, 56, 58, 70 and 82
Population: Results are based on the SAS which included all randomised participants exposed to at least one dose of trial product. "Overall Number of Participants Analyzed" = SAS. "Number Analyzed" = number of participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide 3.0 mg
Number analyzed (Participants) | 125
Participants
  Weeks 0 | 0
  Weeks 30: number analyzed (Participants) | 117
  Weeks 30 | 6
  Weeks 56: number analyzed (Participants) | 103
  Weeks 56 | 5
  Weeks 58: number analyzed (Participants) | 113
  Weeks 58 | 11
  Weeks 70: number analyzed (Participants) | 102
  Weeks 70 | 6
  Weeks 82: number analyzed (Participants) | 100
  Weeks 82 | 2

34. Secondary Outcome: Change in Pulse
Description: Change in pulse was evaluated from baseline (week 0) to weeks 30 and 56, and from week 56 to week 82. Results are based on the participants who completed the corresponding trial period, week 0-30, week 0-56 or week 0-82.
Time Frame: (Week 0, week 30); (Week 0, week 56); (Week 56, week 82)
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: Beats/minute
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 125 | 126
Beats/minute
  Change from week 0 to week 30: number analyzed (Participants) | 116 | 114
  Change from week 0 to week 30 | 4 (12) | -1 (12)
  Change from week 0 to week 56: number analyzed (Participants) | 101 | 101
  Change from week 0 to week 56 | 4 (11) | -1 (12)
  Change from week 56 to week 82: number analyzed (Participants) | 98 | 98
  Change from week 56 to week 82 | -3 (9) | 2 (11)

35. Secondary Outcome: Change in ECG
Description: This outcome measure presents number of subjects with electrocardiogram findings, "normal; abnormal, not clinically significant (NCS) or abnormal, clinically significant (CS)" recorded at baseline (week -14), week 30 and week 56. These findings were categorised by the investigator. Electrocardiogram (ECG) data at week 82 was not collected, thus could not be evaluated. Week 30 and 56 results are based on the participants who completed the corresponding trial period, week 0-30 or week 0-56.
Time Frame: Week -14, week 30, week 56 and week 82
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 125 | 126
Participants
  Week -14: Normal | 102 | 100
  Week -14: Abnormal, NCS | 23 | 26
  Week -14: Abnormal, CS | 0 | 0
  Week 30: number analyzed (Participants) | 117 | 116
  Week 30: Normal | 97 | 95
  Week 30: Abnormal, NCS | 20 | 21
  Week 30: Abnormal, CS | 0 | 0
  Week 56: number analyzed (Participants) | 104 | 103
  Week 56: Normal | 83 | 80
  Week 56: Abnormal, NCS | 21 | 23
  Week 56: Abnormal, CS | 0 | 0
  Week 82: number analyzed (Participants) | 0 | 0

36. Secondary Outcome: Change in Haematology: Haemoglobin
Description: Change in haemoglobin was evaluated from baseline (week 0) to weeks 30 and 56, and from week 56 to week 82. Results are based on the participants who completed the corresponding trial period, week 0-30, week 0-56 or week 0-82.
Time Frame: (Week 0, week 30); (Week 0, week 56); (Week 56, week 82)
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 125 | 126
mmol/L
  Change from week 0 to week 30: number analyzed (Participants) | 114 | 115
  Change from week 0 to week 30 | 0.2 (0.5) | 0.0 (0.4)
  Change from week 0 to week 56: number analyzed (Participants) | 103 | 99
  Change from week 0 to week 56 | 0.3 (0.6) | 0.1 (0.6)
  Change from week 56 to week 82: number analyzed (Participants) | 96 | 92
  Change from week 56 to week 82 | -0.1 (0.6) | -0.0 (0.4)

37. Secondary Outcome: Change in Haematology: Haematocrit
Description: Change in haematocrit was evaluated from baseline (week 0) to weeks 30 and 56, and from week 56 to week 82. Results are based on the participants who completed the corresponding trial period, week 0-30, week 0-56 or week 0-82.
Time Frame: (Week 0, week 30); (Week 0, week 56); (Week 56, week 82)
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: % of red blood cells
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 125 | 126
% of red blood cells
  Change from week 0 to week 30: number analyzed (Participants) | 114 | 114
  Change from week 0 to week 30 | 0.7 (2.3) | 0.1 (2.4)
  Change from week 0 to week 56: number analyzed (Participants) | 103 | 99
  Change from week 0 to week 56 | 1.2 (2.7) | 0.4 (2.8)
  Change from week 56 to week 82: number analyzed (Participants) | 96 | 92
  Change from week 56 to week 82 | -0.4 (2.9) | -0.4 (1.9)

38. Secondary Outcome: Change in Haematology: Thrombocytes, Leucocytes, Eosinophils, Neutrophils, Basophils, Lymphocytes and Monocytes
Description: Change in haematological parameters, "thrombocytes, leucocytes, eosinophils, neutrophils, basophils, lymphocytes and monocytes" was evaluated from baseline (week 0) to weeks 30 and 56, and from week 56 to week 82. Results are based on the participants who completed the corresponding trial period, week 0-30, week 0-56 or week 0-82.
Time Frame: (Week 0, week 30); (Week 0, week 56); (Week 56, week 82)
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 125 | 126
10^9 cells/L
  Thrombocytes: Change from week 0 to week 30: number analyzed (Participants) | 113 | 114
  Thrombocytes: Change from week 0 to week 30 | 9 (37) | 14 (38)
  Thrombocytes: Change from week 0 to week 56: number analyzed (Participants) | 102 | 99
  Thrombocytes: Change from week 0 to week 56 | 7 (46) | 7 (39)
  Thrombocytes: Change from week 56 to week 82: number analyzed (Participants) | 95 | 92
  Thrombocytes: Change from week 56 to week 82 | -2 (31) | 3 (37)
  Leucocytes: Change from week 0 to week 30: number analyzed (Participants) | 114 | 115
  Leucocytes: Change from week 0 to week 30 | 0.1 (1.6) | -0.1 (2)
  Leucocytes: Change from week 0 to week 56: number analyzed (Participants) | 103 | 99
  Leucocytes: Change from week 0 to week 56 | -0.2 (1.6) | -0.4 (1.7)
  Leucocytes: Change from week 56 to week 82: number analyzed (Participants) | 94 | 91
  Leucocytes: Change from week 56 to week 82 | 0.2 (1.5) | 0.0 (2.0)
  Eosinophils: Change from week 0 to week 30: number analyzed (Participants) | 112 | 114
  Eosinophils: Change from week 0 to week 30 | 0.03 (0.15) | 0.04 (0.29)
  Eosinophils: Change from week 0 to week 56: number analyzed (Participants) | 103 | 97
  Eosinophils: Change from week 0 to week 56 | 0.01 (0.15) | 0.00 (0.23)
  Eosinophils: Change from week 56 to week 82: number analyzed (Participants) | 94 | 89
  Eosinophils: Change from week 56 to week 82 | -0.01 (0.12) | 0.00 (0.15)
  Neutrophils: Change from week 0 to week 30: number analyzed (Participants) | 112 | 114
  Neutrophils: Change from week 0 to week 30 | 0.18 (1.33) | -0.01 (1.71)
  Neutrophils: Change from week 0 to week 56: number analyzed (Participants) | 103 | 97
  Neutrophils: Change from week 0 to week 56 | -0.01 (1.49) | -0.13 (1.50)
  Neutrophils: Change from week 56 to week 82: number analyzed (Participants) | 94 | 89
  Neutrophils: Change from week 56 to week 82 | 0.21 (1.35) | -0.00 (1.71)
  Basophils: Change from week 0 to week 30: number analyzed (Participants) | 112 | 114
  Basophils: Change from week 0 to week 30 | 0.01 (0.03) | 0.01 (0.03)
  Basophils: Change from week 0 to week 56: number analyzed (Participants) | 103 | 97
  Basophils: Change from week 0 to week 56 | 0.01 (0.03) | 0.02 (0.03)
  Basophils: Change from week 56 to week 82: number analyzed (Participants) | 94 | 89
  Basophils: Change from week 56 to week 82 | 0.00 (0.03) | 0.00 (0.03)
  Lymphocytes: Change from week 0 to week 30: number analyzed (Participants) | 112 | 114
  Lymphocytes: Change from week 0 to week 30 | -0.18 (0.69) | -0.14 (0.62)
  Lymphocytes: Change from week 0 to week 56: number analyzed (Participants) | 103 | 97
  Lymphocytes: Change from week 0 to week 56 | -0.28 (0.59) | -0.27 (0.72)
  Lymphocytes: Change from week 56 to week 82: number analyzed (Participants) | 94 | 89
  Lymphocytes: Change from week 56 to week 82 | -0.03 (0.48) | -0.00 (0.61)
  Monocytes: Change from week 0 to week 30: number analyzed (Participants) | 112 | 114
  Monocytes: Change from week 0 to week 30 | 0.04 (0.16) | 0.00 (0.18)
  Monocytes: Change from week 0 to week 56: number analyzed (Participants) | 103 | 97
  Monocytes: Change from week 0 to week 56 | 0.06 (0.13) | 0.01 (0.17)
  Monocytes: Change from week 56 to week 82: number analyzed (Participants) | 94 | 89
  Monocytes: Change from week 56 to week 82 | -0.00 (0.15) | 0.04 (0.18)

39. Secondary Outcome: Change in Haematology: Erythrocytes
Description: Change in erythrocytes was evaluated from baseline (week 0) to weeks 30 and 56, and from week 56 to week 82. Results are based on the participants who completed the corresponding trial period, week 0-30, week 0-56 or week 0-82.
Time Frame: (Week 0, week 30); (Week 0, week 56); (Week 56, week 82)
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: 10^12 cells/L
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 125 | 126
10^12 cells/L
  Change from week 0 to week 30: number analyzed (Participants) | 114 | 115
  Change from week 0 to week 30 | 0.0 (0.2) | -0.0 (0.3)
  Change from week 0 to week 56: number analyzed (Participants) | 103 | 99
  Change from week 0 to week 56 | -0.0 (0.3) | -0.1 (0.3)
  Change from week 56 to week 82: number analyzed (Participants) | 96 | 92
  Change from week 56 to week 82 | -0.1 (0.3) | 0.0 (0.2)

40. Secondary Outcome: Change in Biochemistry: Creatinine and Bilirubin (Total)
Description: Change in creatinine and bilirubin (total) was evaluated from baseline (week 0) to weeks 30 and 56, and from week 56 to week 82. Results are based on the participants who completed the corresponding trial period, week 0-30, week 0-56 or week 0-82.
Time Frame: (Week 0, week 30); (Week 0, week 56); (Week 56, week 82)
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 125 | 126
umol/L
  Creatinine: Change from week 0 to week 30: number analyzed (Participants) | 116 | 116
  Creatinine: Change from week 0 to week 30 | 1 (7) | 0 (8)
  Creatinine: Change from week 0 to week 56: number analyzed (Participants) | 105 | 101
  Creatinine: Change from week 0 to week 56 | 2 (7) | 4 (9)
  Creatinine: Change from week 56 to week 82: number analyzed (Participants) | 99 | 97
  Creatinine: Change from week 56 to week 82 | 2 (8) | 1 (10)
  Bilirubin (total): Change from week 0 to week 30: number analyzed (Participants) | 116 | 114
  Bilirubin (total): Change from week 0 to week 30 | 1 (4) | 1 (5)
  Bilirubin (total): Change from week 0 to week 56: number analyzed (Participants) | 105 | 101
  Bilirubin (total): Change from week 0 to week 56 | 1 (4) | 1 (5)
  Bilirubin (total): Change from week 56 to week 82: number analyzed (Participants) | 99 | 96
  Bilirubin (total): Change from week 56 to week 82 | 0 (5) | -0 (4)

41. Secondary Outcome: Change in Biochemistry: Creatinine Kinase, Amylase, Lipase, ALT, AST and ALP
Description: Change in biochemistry parameters, "creatinine kinase, amylase, lipase, alanine aminotransferase (ALT), aspartate aminotransferase (AST) and alkaline phosphatase (ALP)" was evaluated from baseline (week 0) to weeks 30 and 56, and from week 56 to week 82. Results are based on the participants who completed the corresponding trial period, week 0-30, week 0-56 or week 0-82.
Time Frame: (Week 0, week 30); (Week 0, week 56); (Week 56, week 82)
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 125 | 126
U/L
  Creatinine kinase: Change from week 0 to week 30: number analyzed (Participants) | 116 | 116
  Creatinine kinase: Change from week 0 to week 30 | 13 (251) | 0 (225)
  Creatinine kinase: Change from week 0 to week 56: number analyzed (Participants) | 105 | 101
  Creatinine kinase: Change from week 0 to week 56 | 32 (228) | 0 (111)
  Creatinine kinase: Change from week 56 to week 82: number analyzed (Participants) | 99 | 97
  Creatinine kinase: Change from week 56 to week 82 | 28 (321) | 4 (114)
  Amylase: Change from week 0 to week 30: number analyzed (Participants) | 116 | 116
  Amylase: Change from week 0 to week 30 | 4 (12) | 3 (16)
  Amylase: Change from week 0 to week 56: number analyzed (Participants) | 105 | 101
  Amylase: Change from week 0 to week 56 | 2 (10) | -0 (9)
  Amylase: Change from week 56 to week 82: number analyzed (Participants) | 99 | 97
  Amylase: Change from week 56 to week 82 | -1 (8) | 1 (11)
  Lipase: Change from week 0 to week 30: number analyzed (Participants) | 116 | 116
  Lipase: Change from week 0 to week 30 | 6 (13) | 1 (19)
  Lipase: Change from week 0 to week 56: number analyzed (Participants) | 105 | 101
  Lipase: Change from week 0 to week 56 | 3 (13) | -2 (5)
  Lipase: Change from week 56 to week 82: number analyzed (Participants) | 99 | 97
  Lipase: Change from week 56 to week 82 | -4 (9) | -0 (5)
  ALT: Change from week 0 to week 30: number analyzed (Participants) | 116 | 116
  ALT: Change from week 0 to week 30 | -2 (15) | -1 (15)
  ALT: Change from week 0 to week 56: number analyzed (Participants) | 105 | 101
  ALT: Change from week 0 to week 56 | -2 (16) | -0 (23)
  ALT: Change from week 56 to week 82: number analyzed (Participants) | 99 | 97
  ALT: Change from week 56 to week 82 | 1 (12) | 2 (20)
  AST: Change from week 0 to week 30: number analyzed (Participants) | 116 | 116
  AST: Change from week 0 to week 30 | -1 (8) | -1 (11)
  AST: Change from week 0 to week 56: number analyzed (Participants) | 105 | 101
  AST: Change from week 0 to week 56 | -1 (8) | -1 (11)
  AST: Change from week 56 to week 82: number analyzed (Participants) | 99 | 97
  AST: Change from week 56 to week 82 | 1 (12) | 1 (11)
  ALP: Change from week 0 to week 30: number analyzed (Participants) | 116 | 116
  ALP: Change from week 0 to week 30 | -16 (25) | -8 (66)
  ALP: Change from week 0 to week 56: number analyzed (Participants) | 105 | 101
  ALP: Change from week 0 to week 56 | -23 (36) | -19 (53)
  ALP: Change from week 56 to week 82: number analyzed (Participants) | 99 | 97
  ALP: Change from week 56 to week 82 | -2 (22) | -10 (24)

42. Secondary Outcome: Change in Biochemistry: Urea (BUN), Sodium, Potassium, Calcium Total and Calcium Albumin-corrected
Description: Change in biochemistry parameters, "urea (blood urea nitrogen [BUN]), sodium, potassium, calcium total and calcium (Ca) albumin-corrected" was evaluated from baseline (week [Wk] 0) to weeks 30 and 56, and from week 56 to week 82. Results are based on the participants who completed the corresponding trial period, week 0-30, week 0-56 or week 0-82.
Time Frame: (Week 0, week 30); (Week 0, week 56); (Week 56, week 82)
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 125 | 126
mmol/L
  Urea (BUN): Change from week 0 to week 30: number analyzed (Participants) | 116 | 116
  Urea (BUN): Change from week 0 to week 30 | -0.06 (1.07) | 0.00 (1.14)
  Urea (BUN): Change from week 0 to week 56: number analyzed (Participants) | 105 | 101
  Urea (BUN): Change from week 0 to week 56 | -0.26 (1.01) | -0.05 (1.19)
  Urea (BUN): Change from week 56 to week 82: number analyzed (Participants) | 99 | 97
  Urea (BUN): Change from week 56 to week 82 | 0.23 (1.11) | 0.00 (1.07)
  Sodium: Change from week 0 to week 30: number analyzed (Participants) | 116 | 116
  Sodium: Change from week 0 to week 30 | 0 (2) | 0 (2)
  Sodium: Change from week 0 to week 56: number analyzed (Participants) | 105 | 101
  Sodium: Change from week 0 to week 56 | 0 (2) | 0 (3)
  Sodium: Change from week 56 to week 82: number analyzed (Participants) | 99 | 97
  Sodium: Change from week 56 to week 82 | -1 (3) | -1 (3)
  Potassium: Change from week 0 to week 30: number analyzed (Participants) | 116 | 116
  Potassium: Change from week 0 to week 30 | -0.0 (0.4) | 0.0 (0.3)
  Potassium: Change from week 0 to week 56: number analyzed (Participants) | 105 | 101
  Potassium: Change from week 0 to week 56 | -0.1 (0.4) | -0.0 (0.3)
  Potassium: Change from week 56 to week 82: number analyzed (Participants) | 99 | 97
  Potassium: Change from week 56 to week 82 | 0.0 (0.3) | -0.0 (0.4)
  Calcium total: Change from week 0 to week 30: number analyzed (Participants) | 116 | 116
  Calcium total: Change from week 0 to week 30 | -0.01 (0.09) | -0.03 (0.09)
  Calcium total: Change from week 0 to week 56: number analyzed (Participants) | 105 | 101
  Calcium total: Change from week 0 to week 56 | -0.04 (0.10) | -0.04 (0.09)
  Calcium total: Change from week 56 to week 82: number analyzed (Participants) | 99 | 97
  Calcium total: Change from week 56 to week 82 | -0.00 (0.09) | -0.01 (0.09)
  Ca albumin-corrected:Change from week 0 to week 30: number analyzed (Participants) | 116 | 116
  Ca albumin-corrected:Change from week 0 to week 30 | -0.04 (0.09) | -0.03 (0.09)
  Ca albumin-corrected:Change from week 0 to week 56: number analyzed (Participants) | 105 | 101
  Ca albumin-corrected:Change from week 0 to week 56 | -0.07 (0.10) | -0.07 (0.08)
  Ca albumin-corrected: Change from Wk 56 to Wk 82: number analyzed (Participants) | 99 | 97
  Ca albumin-corrected: Change from Wk 56 to Wk 82 | 0.01 (0.07) | -0.00 (0.09)

43. Secondary Outcome: Change in Biochemistry: Albumin
Description: Change in albumin was evaluated from baseline (week 0) to weeks 30 and 56, and from week 56 to week 82. Results are based on the participants who completed the corresponding trial period, week 0-30, week 0-56 or week 0-82.
Time Frame: (Week 0, week 30); (Week 0, week 56); (Week 56, week 82)
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 125 | 126
g/dL
  Change from week 0 to week 30: number analyzed (Participants) | 116 | 116
  Change from week 0 to week 30 | 0.1 (0.2) | 0.0 (0.3)
  Change from week 0 to week 56: number analyzed (Participants) | 105 | 101
  Change from week 0 to week 56 | 0.1 (0.3) | 0.1 (0.3)
  Change from week 56 to week 82: number analyzed (Participants) | 99 | 97
  Change from week 56 to week 82 | -0.0 (0.2) | -0.0 (0.3)

44. Secondary Outcome: Change in Biochemistry: CEA
Description: Change in carcinoembryonic antigen (CEA) was evaluated from baseline (week 0) to weeks 30 and 56, and from week 56 to week 82. Results are based on the participants who completed the corresponding trial period, week 0-30, week 0-56 or week 0-82.
Time Frame: (Week 0, week 30); (Week 0, week 56); (Week 56, week 82)
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 125 | 126
ng/mL
  Change from week 0 to week 30: number analyzed (Participants) | 116 | 115
  Change from week 0 to week 30 | -0.0 (0.3) | -0.1 (0.6)
  Change from week 0 to week 56: number analyzed (Participants) | 104 | 101
  Change from week 0 to week 56 | 0.0 (0.4) | -0.0 (0.6)
  Change from week 56 to week 82: number analyzed (Participants) | 98 | 96
  Change from week 56 to week 82 | 0.0 (0.4) | 0.0 (0.3)

45. Secondary Outcome: Change in Hormone Level: Calcitonin
Description: Change in calcitonin was evaluated from baseline (week 0) to weeks 30 and 56, and from week 56 to week 82. Results are based on the participants who completed the corresponding trial period, week 0-30, week 0-56 or week 0-82.
Time Frame: (Week 0, week 30); (Week 0, week 56); (Week 56, week 82)
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 125 | 126
ng/L
  Change from week 0 to week 30: number analyzed (Participants) | 116 | 113
  Change from week 0 to week 30 | 0.1 (0.8) | 0.1 (0.7)
  Change from week 0 to week 56: number analyzed (Participants) | 105 | 99
  Change from week 0 to week 56 | 0.0 (0.7) | -0.0 (0.8)
  Change from week 56 to week 82: number analyzed (Participants) | 99 | 94
  Change from week 56 to week 82 | -0.1 (0.6) | 0.2 (1.5)

46. Secondary Outcome: Change in Hormone Level: TSH and Prolactin
Description: Change in hormone levels, "thyroid stimulating hormone (TSH) and prolactin" was evaluated from baseline (week 0) to weeks 30 and 56, and from week 56 to week 82. Results are based on the participants who completed the corresponding trial period, week 0-30, week 0-56 or week 0-82.
Time Frame: (Week 0, week 30); (Week 0, week 56); (Week 56, week 82)
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: mIU/L
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 125 | 126
mIU/L
  TSH: Change from week 0 to week 30: number analyzed (Participants) | 115 | 114
  TSH: Change from week 0 to week 30 | -0.35 (1.37) | -0.08 (1.17)
  TSH: Change from week 0 to week 56: number analyzed (Participants) | 104 | 99
  TSH: Change from week 0 to week 56 | -0.42 (1.36) | -0.14 (1.28)
  TSH: Change from week 56 to week 82: number analyzed (Participants) | 96 | 97
  TSH: Change from week 56 to week 82 | 0.38 (1.91) | 0.13 (1.57)
  Prolactin: Change from week 0 to week 30: number analyzed (Participants) | 115 | 116
  Prolactin: Change from week 0 to week 30 | 23 (165) | -47 (452)
  Prolactin: Change from week 0 to week 56: number analyzed (Participants) | 104 | 101
  Prolactin: Change from week 0 to week 56 | 63 (312) | -63 (684)
  Prolactin: Change from week 56 to week 82: number analyzed (Participants) | 98 | 97
  Prolactin: Change from week 56 to week 82 | -29 (396) | 13 (98)

47. Secondary Outcome: Change in Hormone Level: Free T4 and ACTH
Description: Change in hormone levels, "thyroxine (T4) and adrenocorticotropic hormone (ACTH)" was evaluated from baseline (week 0) to weeks 30 and 56, and from week 56 to week 82. Results are based on the participants who completed the corresponding trial period, week 0-30, week 0-56 or week 0-82.
Time Frame: (Week 0, week 30); (Week 0, week 56); (Week 56, week 82)
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 125 | 126
pmol/L
  T4: Change from week 0 to week 30: number analyzed (Participants) | 115 | 116
  T4: Change from week 0 to week 30 | 0.6 (1.9) | 0.8 (2.1)
  T4: Change from week 0 to week 56: number analyzed (Participants) | 104 | 101
  T4: Change from week 0 to week 56 | 0.3 (1.8) | 0.6 (2.1)
  T4: Change from week 56 to week 82: number analyzed (Participants) | 98 | 97
  T4: Change from week 56 to week 82 | 0.0 (1.6) | 0.2 (2.3)
  ACTH: Change from week 0 to week 30: number analyzed (Participants) | 111 | 113
  ACTH: Change from week 0 to week 30 | 0.4 (4.4) | 0.5 (3.9)
  ACTH: Change from week 0 to week 56: number analyzed (Participants) | 100 | 100
  ACTH: Change from week 0 to week 56 | 0.6 (4.9) | 0.6 (3.8)
  ACTH: Change from week 56 to week 82: number analyzed (Participants) | 98 | 96
  ACTH: Change from week 56 to week 82 | -0.8 (4.7) | -0.4 (2.9)

48. Secondary Outcome: Change in Hormone Level: IGF-1 and Cortisol
Description: Change in hormone levels, "insulin-like growth factor-1 (IGF-1) and cortisol" was evaluated from baseline (week 0) to weeks 30 and 56, and from week 56 to week 82. Results are based on the participants who completed the corresponding trial period, week 0-30, week 0-56 or week 0-82.
Time Frame: (Week 0, week 30); (Week 0, week 56); (Week 56, week 82)
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 125 | 126
ng/mL
  IGF-1: Change from week 0 to week 30: number analyzed (Participants) | 116 | 114
  IGF-1: Change from week 0 to week 30 | 10.61 (89.83) | 3.79 (101.12)
  IGF-1: Change from week 0 to week 56: number analyzed (Participants) | 105 | 101
  IGF-1: Change from week 0 to week 56 | -4.60 (84.51) | 3.69 (111.63)
  IGF-1: Change from week 56 to week 82: number analyzed (Participants) | 99 | 96
  IGF-1: Change from week 56 to week 82 | -14.60 (80.82) | -16.35 (65.89)
  Cortisol: Change from week 0 to week 30: number analyzed (Participants) | 115 | 116
  Cortisol: Change from week 0 to week 30 | 6.9 (66.9) | 8.6 (60.1)
  Cortisol: Change from week 0 to week 56: number analyzed (Participants) | 104 | 101
  Cortisol: Change from week 0 to week 56 | 5.1 (65.2) | 8.5 (57.9)
  Cortisol: Change from week 56 to week 82: number analyzed (Participants) | 97 | 97
  Cortisol: Change from week 56 to week 82 | 0.6 (66.6) | 10.4 (61.2)

49. Secondary Outcome: Change in Hormone Level: DHEAS
Description: Change in dehydroepiandrosterone sulfate (DHEAS) was evaluated from baseline (week 0) to weeks 30 and 56, and from week 56 to week 82. Results are based on the participants who completed the corresponding trial period, week 0-30, week 0-56 or week 0-82.
Time Frame: (Week 0, week 30); (Week 0, week 56); (Week 56, week 82)
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 125 | 126
umol/L
  Change from week 0 to week 30: number analyzed (Participants) | 116 | 114
  Change from week 0 to week 30 | 0.94 (1.66) | 0.57 (1.78)
  Change from week 0 to week 56: number analyzed (Participants) | 103 | 101
  Change from week 0 to week 56 | 0.95 (1.91) | 0.89 (2.05)
  Change from week 56 to week 82: number analyzed (Participants) | 97 | 97
  Change from week 56 to week 82 | -0.08 (2.11) | -0.05 (1.27)

50. Secondary Outcome: Change in Hormone Level: LH and FSH
Description: Change in hormone levels, "luteinising hormone (LH) and follicle stimulating hormone (FSH)" was evaluated from baseline (week 0) to weeks 30 and 56, and from week 56 to week 82. Results are based on the participants who completed the corresponding trial period, week 0-30, week 0-56 or week 0-82.
Time Frame: (Week 0, week 30); (Week 0, week 56); (Week 56, week 82)
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 125 | 126
IU/L
  LH: Change from week 0 to week 30: number analyzed (Participants) | 115 | 116
  LH: Change from week 0 to week 30 | 0.4 (9.1) | 0.7 (7.9)
  LH: Change from week 0 to week 56: number analyzed (Participants) | 104 | 101
  LH: Change from week 0 to week 56 | 0.2 (9.1) | 0.6 (6.6)
  LH: Change from week 56 to week 82: number analyzed (Participants) | 98 | 97
  LH: Change from week 56 to week 82 | 0.4 (8.7) | -0.5 (8.0)
  FSH: Change from week 0 to week 30: number analyzed (Participants) | 113 | 114
  FSH: Change from week 0 to week 30 | 0.2 (2.6) | -0.2 (2.7)
  FSH: Change from week 0 to week 56: number analyzed (Participants) | 104 | 98
  FSH: Change from week 0 to week 56 | 0.6 (4.0) | 0.1 (2.5)
  FSH: Change from week 56 to week 82: number analyzed (Participants) | 96 | 96
  FSH: Change from week 56 to week 82 | -0.1 (3.6) | -0.1 (3.1)

51. Secondary Outcome: Change in Hormone Level: Estradiol (Females)
Description: Change in estradiol (only for female) was evaluated from baseline (week 0) to weeks 30 and 56, and from week 56 to week 82. Results are based on the participants who completed the corresponding trial period, week 0-30, week 0-56 or week 0-82.
Time Frame: (Week 0, week 30); (Week 0, week 56); (Week 56, week 82)
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 71 | 78
pg/mL
  Change from week 0 to week 30: number analyzed (Participants) | 65 | 71
  Change from week 0 to week 30 | -5.0 (81.0) | 20.2 (67.6)
  Change from week 0 to week 56: number analyzed (Participants) | 56 | 60
  Change from week 0 to week 56 | 11.6 (94.4) | 14.1 (63.6)
  Change from week 56 to week 82: number analyzed (Participants) | 52 | 58
  Change from week 56 to week 82 | -2.3 (89.1) | -1.7 (65.3)

52. Secondary Outcome: Change in Hormone Level: Testosterone (Males)
Description: This outcome measure presents "testosterone (only for males) results" for baseline (week 0), week 30, week 56 and week 82. ADVIA Centaur Testosterone (TSTO) assay was used for the evaluation of testosterone hormone. Week 30, 56 and 82 results are based on the participants who completed the corresponding trial period, week 0-30, week 0-56 or week 0-82.
Time Frame: Week 0, week 30, week 56 and week 82
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 54 | 48
nmol/L
  Week 0: number analyzed (Participants) | 53 | 48
  Week 0 | 8.13 (3.45) | 8.06 (3.66)
  Week 30: number analyzed (Participants) | 51 | 45
  Week 30 | 10.00 (4.02) | 9.33 (5.27)
  Week 56: number analyzed (Participants) | 39 | 33
  Week 56 | 10.55 (4.14) | 9.51 (3.31)
  Week 82: number analyzed (Participants) | 9 | 5
  Week 82 | 11.36 (5.27) | 6.16 (3.27)

53. Secondary Outcome: Change in NTX1
Description: Change in type I collagen N-telopeptide (NTX1) was evaluated from baseline (week 0) to weeks 30 and 56, and from week 56 to week 82. Results are presented in "nmol bone collagen equivalents (BCE)/L". Results are based on the participants who completed the corresponding trial period, week 0-30, week 0-56 or week 0-82.
Time Frame: (Week 0, week 30); (Week 0, week 56); (Week 56, week 82)
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: nmol BCE/L
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 125 | 126
nmol BCE/L
  Change from week 0 to week 30: number analyzed (Participants) | 116 | 114
  Change from week 0 to week 30 | -2.4 (10.4) | -3.2 (12.0)
  Change from week 0 to week 56: number analyzed (Participants) | 104 | 101
  Change from week 0 to week 56 | -3.7 (14.1) | -2.9 (15.1)
  Change from week 56 to week 82: number analyzed (Participants) | 97 | 97
  Change from week 56 to week 82 | -2.8 (12.8) | -4.6 (10.0)

54. Secondary Outcome: Change in CTX1
Description: Change in type I collagen C-telopeptide (CTX1) was evaluated from baseline (week 0) to weeks 30 and 56, and from week 56 to week 82. Results are based on the participants who completed the corresponding trial period, week 0-30, week 0-56 or week 0-82.
Time Frame: (Week 0, week 30); (Week 0, week 56); (Week 56, week 82)
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 125 | 126
pg/mL
  Change from week 0 to week 30: number analyzed (Participants) | 115 | 114
  Change from week 0 to week 30 | -7 (358) | -84 (404)
  Change from week 0 to week 56: number analyzed (Participants) | 104 | 100
  Change from week 0 to week 56 | -36 (353) | -97 (473)
  Change from week 56 to week 82: number analyzed (Participants) | 99 | 97
  Change from week 56 to week 82 | -107 (359) | -162 (318)

55. Secondary Outcome: Change in P1NP
Description: Change in procollagen 1 N-terminal propeptide (P1NP) was evaluated from baseline (week 0) to weeks 30 and 56, and from week 56 to week 82. Results are based on the participants who completed the corresponding trial period, week 0-30, week 0-56 or week 0-82.
Time Frame: (Week 0, week 30); (Week 0, week 56); (Week 56, week 82)
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 125 | 126
ng/mL
  Change from week 0 to week 30: number analyzed (Participants) | 115 | 115
  Change from week 0 to week 30 | -35 (124) | -30 (184)
  Change from week 0 to week 56: number analyzed (Participants) | 105 | 101
  Change from week 0 to week 56 | -55 (151) | -63 (192)
  Change from week 56 to week 82: number analyzed (Participants) | 99 | 95
  Change from week 56 to week 82 | -30 (107) | -47 (84)

56. Secondary Outcome: Change in Alkaline Phosphatase (Bone)
Description: Change in alkaline phosphatase (bone specific) was evaluated from baseline (week 0) to weeks 30 and 56, and from week 56 to week 82. Results are based on the participants who completed the corresponding trial period, week 0-30, week 0-56 or week 0-82.
Time Frame: (Week 0, week 30); (Week 0, week 56); (Week 56, week 82)
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 125 | 126
U/L
  Change from week 0 to week 30: number analyzed (Participants) | 116 | 113
  Change from week 0 to week 30 | -15 (16) | -12 (26)
  Change from week 0 to week 56: number analyzed (Participants) | 105 | 100
  Change from week 0 to week 56 | -17 (18) | -17 (30)
  Change from week 56 to week 82: number analyzed (Participants) | 99 | 96
  Change from week 56 to week 82 | -1 (11) | -4 (12)

57. Secondary Outcome: Change in Pubertal Status
Description: This outcome measure presents "pubertal status results" which is based on Tanner staging (Tanner stage 2-5), recorded at baseline (week 0), week 30, week 56 and week 82. Results are presented for the following categories: 1) For female: breast development and pubic hair development (by Tanner staging). 2) For male: penis development and pubic hair development (by Tanner staging). Each category shows number of participants in stages 2 to 5, where stage 2 represents "early pubertal development" and stage 5 represents "pubertal development equivalent to that of an adult". Week 30, 56 and 82 results are based on the participants who completed the corresponding trial period, week 0-30, week 0-56 or week 0-82.
Time Frame: (Week 0, week 30); (Week 0, week 56); (Week 56, week 82)
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 125 | 126
Participants
  Week 0: Breast development (for female): number analyzed (Participants) | 71 | 78
  Week 0: Breast development (for female): Stage 2 | 2 | 1
  Week 0: Breast development (for female): Stage 3 | 6 | 8
  Week 0: Breast development (for female): Stage 4 | 23 | 30
  Week 0: Breast development (for female): Stage 5 | 40 | 39
  Week 30: Breast development (for female): number analyzed (Participants) | 66 | 74
  Week 30: Breast development (for female): Stage 2 | 1 | 0
  Week 30: Breast development (for female): Stage 3 | 4 | 6
  Week 30: Breast development (for female): Stage 4 | 22 | 25
  Week 30: Breast development (for female): Stage 5 | 39 | 43
  Week 56: Breast development (for female): number analyzed (Participants) | 57 | 63
  Week 56: Breast development (for female): Stage 2 | 0 | 0
  Week 56: Breast development (for female): Stage 3 | 2 | 2
  Week 56: Breast development (for female): Stage 4 | 14 | 20
  Week 56: Breast development (for female): Stage 5 | 41 | 41
  Week 82: Breast development (for female): number analyzed (Participants) | 53 | 61
  Week 82: Breast development (for female): Stage 2 | 0 | 0
  Week 82: Breast development (for female): Stage 3 | 0 | 2
  Week 82: Breast development (for female): Stage 4 | 7 | 13
  Week 82: Breast development (for female): Stage 5 | 46 | 46
  Week 0: Pubic hair development (for female): number analyzed (Participants) | 71 | 78
  Week 0: Pubic hair development (for female): Stage 2 | 2 | 3
  Week 0: Pubic hair development (for female): Stage 3 | 6 | 5
  Week 0: Pubic hair development (for female): Stage 4 | 22 | 26
  Week 0: Pubic hair development (for female): Stage 5 | 41 | 44
  Week 30: Pubic hair development (for female): number analyzed (Participants) | 66 | 74
  Week 30: Pubic hair development (for female): Stage 2 | 1 | 0
  Week 30: Pubic hair development (for female): Stage 3 | 4 | 4
  Week 30: Pubic hair development (for female): Stage 4 | 20 | 25
  Week 30: Pubic hair development (for female): Stage 5 | 41 | 45
  Week 56: Pubic hair development (for female): number analyzed (Participants) | 57 | 63
  Week 56: Pubic hair development (for female): Stage 2 | 1 | 0
  Week 56: Pubic hair development (for female): Stage 3 | 2 | 2
  Week 56: Pubic hair development (for female): Stage 4 | 13 | 21
  Week 56: Pubic hair development (for female): Stage 5 | 41 | 40
  Week 82: Pubic hair development (for female): number analyzed (Participants) | 53 | 61
  Week 82: Pubic hair development (for female): Stage 2 | 0 | 0
  Week 82: Pubic hair development (for female): Stage 3 | 1 | 2
  Week 82: Pubic hair development (for female): Stage 4 | 7 | 14
  Week 82: Pubic hair development (for female): Stage 5 | 45 | 45
  Week 0: penis development (male): number analyzed (Participants) | 54 | 48
  Week 0: penis development (male): Stage 2 | 4 | 7
  Week 0: penis development (male): Stage 3 | 11 | 8
  Week 0: penis development (male): Stage 4 | 16 | 14
  Week 0: penis development (male): Stage 5 | 23 | 19
  Week 30: penis development (male): number analyzed (Participants) | 51 | 45
  Week 30: penis development (male): Stage 2 | 1 | 2
  Week 30: penis development (male): Stage 3 | 11 | 7
  Week 30: penis development (male): Stage 4 | 14 | 11
  Week 30: penis development (male): Stage 5 | 25 | 25
  Week 56: penis development (male): number analyzed (Participants) | 48 | 41
  Week 56: penis development (male): Stage 2 | 1 | 0
  Week 56: penis development (male): Stage 3 | 6 | 6
  Week 56: penis development (male): Stage 4 | 15 | 6
  Week 56: penis development (male): Stage 5 | 26 | 29
  Week 82: penis development (male): number analyzed (Participants) | 45 | 38
  Week 82: penis development (male): Stage 2 | 0 | 0
  Week 82: penis development (male): Stage 3 | 3 | 3
  Week 82: penis development (male): Stage 4 | 11 | 6
  Week 82: penis development (male): Stage 5 | 31 | 29
  Week 0: Pubic hair development (male): number analyzed (Participants) | 54 | 48
  Week 0: Pubic hair development (male): Stage 2 | 6 | 9
  Week 0: Pubic hair development (male): Stage 3 | 8 | 5
  Week 0: Pubic hair development (male): Stage 4 | 19 | 13
  Week 0: Pubic hair development (male): Stage 5 | 21 | 21
  Week 30: Pubic hair development (male): number analyzed (Participants) | 50 | 45
  Week 30: Pubic hair development (male): Stage 2 | 1 | 3
  Week 30: Pubic hair development (male): Stage 3 | 10 | 7
  Week 30: Pubic hair development (male): Stage 4 | 15 | 9
  Week 30: Pubic hair development (male): Stage 5 | 24 | 26
  Week 56: Pubic hair development (male): number analyzed (Participants) | 47 | 41
  Week 56: Pubic hair development (male): Stage 2 | 1 | 0
  Week 56: Pubic hair development (male): Stage 3 | 7 | 6
  Week 56: Pubic hair development (male): Stage 4 | 15 | 7
  Week 56: Pubic hair development (male): Stage 5 | 24 | 28
  Week 82: Pubic hair development (male): number analyzed (Participants) | 43 | 38
  Week 82: Pubic hair development (male): Stage 2 | 0 | 0
  Week 82: Pubic hair development (male): Stage 3 | 3 | 2
  Week 82: Pubic hair development (male): Stage 4 | 10 | 8
  Week 82: Pubic hair development (male): Stage 5 | 30 | 28

58. Secondary Outcome: Change in Physical Examination
Description: This outcome measure presents number of subjects with physical examination findings, "normal; abnormal, not clinically significant (NCS) or abnormal, clinically significant (CS)" at baseline (week 0), week 30, week 56 and week 82. These findings were categorised by the investigator. Results include examination of: "general appearance"; "head, ears, eyes, nose, throat, neck"; "respiratory system"; "cardiovascular system (CVS)"; "gastrointestinal (GI) system including mouth"; "musculoskeletal system"; "central nervous system (CNS) and peripheral nervous system (PNS)"; "skin"; "thyroid gland" and "lymph node palpation". Week 30, 56 and 82 results are based on the participants who completed the corresponding trial period, week 0-30, week 0-56 or week 0-82.
Time Frame: Week 0, week 30, week 56 and week 82
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 125 | 126
Participants
  General Appearance: Week 0: Normal | 93 | 101
  General Appearance: Week 0: Abnormal, NCS | 30 | 23
  General Appearance: Week 0: Abnormal, CS | 2 | 2
  General Appearance: Week 30: number analyzed (Participants) | 116 | 116
  General Appearance: Week 30: Normal | 94 | 95
  General Appearance: Week 30: Abnormal, NCS | 21 | 20
  General Appearance: Week 30: Abnormal, CS | 1 | 1
  General Appearance: Week 56: number analyzed (Participants) | 104 | 102
  General Appearance: Week 56: Normal | 84 | 85
  General Appearance: Week 56: Abnormal, NCS | 18 | 16
  General Appearance: Week 56: Abnormal, CS | 2 | 1
  General Appearance: Week 82: number analyzed (Participants) | 99 | 99
  General Appearance: Week 82: Normal | 80 | 81
  General Appearance: Week 82: Abnormal, NCS | 18 | 17
  General Appearance: Week 82: Abnormal, CS | 1 | 1
  Head, ears, eyes, nose, throat, neck: Week 0: Normal | 120 | 116
  Head, ears, eyes, nose, throat, neck: Week 0: Abnormal, NCS | 5 | 10
  Head, ears, eyes, nose, throat, neck: Week 0: Abnormal, CS | 0 | 0
  Head, ears, eyes, nose, throat, neck: Week 30: number analyzed (Participants) | 116 | 116
  Head, ears, eyes, nose, throat, neck: Week 30: Normal | 114 | 107
  Head, ears, eyes, nose, throat, neck: Week 30: Abnormal, NCS | 2 | 9
  Head, ears, eyes, nose, throat, neck: Week 30: Abnormal, CS | 0 | 0
  Head, ears, eyes, nose, throat, neck: Week 56: number analyzed (Participants) | 104 | 102
  Head, ears, eyes, nose, throat, neck: Week 56: Normal | 101 | 98
  Head, ears, eyes, nose, throat, neck: Week 56: Abnormal, NCS | 3 | 4
  Head, ears, eyes, nose, throat, neck: Week 56: Abnormal, CS | 0 | 0
  Head, ears, eyes, nose, throat, neck: Week 82: number analyzed (Participants) | 99 | 99
  Head, ears, eyes, nose, throat, neck: Week 82: Normal | 98 | 94
  Head, ears, eyes, nose, throat, neck: Week 82: Abnormal, NCS | 1 | 5
  Head, ears, eyes, nose, throat, neck: Week 82: Abnormal, CS | 0 | 0
  Respiratory system: Week 0: Normal | 125 | 123
  Respiratory system: Week 0: Abnormal, NCS | 0 | 3
  Respiratory system: Week 0: Abnormal, CS | 0 | 0
  Respiratory system: Week 30: number analyzed (Participants) | 116 | 116
  Respiratory system: Week 30: Normal | 116 | 115
  Respiratory system: Week 30: Abnormal, NCS | 0 | 1
  Respiratory system: Week 30: Abnormal, CS | 0 | 0
  Respiratory system: Week 56: number analyzed (Participants) | 104 | 102
  Respiratory system: Week 56: Normal | 104 | 101
  Respiratory system: Week 56: Abnormal, NCS | 0 | 1
  Respiratory system: Week 56: Abnormal, CS | 0 | 0
  Respiratory system: Week 82: number analyzed (Participants) | 99 | 99
  Respiratory system: Week 82: Normal | 99 | 96
  Respiratory system: Week 82: Abnormal, NCS | 0 | 3
  Respiratory system: Week 82: Abnormal, CS | 0 | 0
  Cardiovascular system: Week 0: Normal | 124 | 125
  Cardiovascular system: Week 0: Abnormal, NCS | 1 | 1
  Cardiovascular system: Week 0: Abnormal, CS | 0 | 0
  Cardiovascular system: Week 30: number analyzed (Participants) | 116 | 116
  Cardiovascular system: Week 30: Normal | 115 | 112
  Cardiovascular system: Week 30: Abnormal, NCS | 1 | 4
  Cardiovascular system: Week 30: Abnormal, CS | 0 | 0
  Cardiovascular system: Week 56: number analyzed (Participants) | 104 | 102
  Cardiovascular system: Week 56: Normal | 102 | 100
  Cardiovascular system: Week 56: Abnormal, NCS | 2 | 2
  Cardiovascular system: Week 56: Abnormal, CS | 0 | 0
  Cardiovascular system: Week 82: number analyzed (Participants) | 99 | 99
  Cardiovascular system: Week 82: Normal | 97 | 98
  Cardiovascular system: Week 82: Abnormal, NCS | 2 | 1
  Cardiovascular system: Week 82: Abnormal, CS | 0 | 0
  GI system including mouth: Week 0: Normal | 119 | 119
  GI system including mouth: Week 0: Abnormal, NCS | 5 | 6
  GI system including mouth: Week 0: Abnormal, CS | 1 | 1
  GI system including mouth: Week 30: number analyzed (Participants) | 116 | 116
  GI system including mouth: Week 30: Normal | 111 | 109
  GI system including mouth: Week 30: Abnormal, NCS | 5 | 6
  GI system including mouth: Week 30: Abnormal, CS | 0 | 1
  GI system including mouth: Week 56: number analyzed (Participants) | 104 | 102
  GI system including mouth: Week 56: Normal | 102 | 98
  GI system including mouth: Week 56: Abnormal, NCS | 2 | 4
  GI system including mouth: Week 56: Abnormal, CS | 0 | 0
  GI system including mouth: Week 82: number analyzed (Participants) | 99 | 99
  GI system including mouth: Week 82: Normal | 96 | 94
  GI system including mouth: Week 82: Abnormal, NCS | 1 | 5
  GI system including mouth: Week 82: Abnormal, CS | 2 | 0
  Musculoskeletal system: Week 0: Normal | 121 | 119
  Musculoskeletal system: Week 0: Abnormal, NCS | 4 | 7
  Musculoskeletal system: Week 0: Abnormal, CS | 0 | 0
  Musculoskeletal system: Week 30: number analyzed (Participants) | 116 | 116
  Musculoskeletal system: Week 30: Normal | 113 | 106
  Musculoskeletal system: Week 30: Abnormal, NCS | 3 | 10
  Musculoskeletal system: Week 30: Abnormal, CS | 0 | 0
  Musculoskeletal system: Week 56: number analyzed (Participants) | 104 | 102
  Musculoskeletal system: Week 56: Normal | 102 | 97
  Musculoskeletal system: Week 56: Abnormal, NCS | 1 | 5
  Musculoskeletal system: Week 56: Abnormal, CS | 1 | 0
  Musculoskeletal system: Week 82: number analyzed (Participants) | 99 | 99
  Musculoskeletal system: Week 82: Normal | 97 | 92
  Musculoskeletal system: Week 82: Abnormal, NCS | 1 | 7
  Musculoskeletal system: Week 82: Abnormal, CS | 1 | 0
  CNS and PNS: Week 0: Normal | 124 | 124
  CNS and PNS: Week 0: Abnormal, NCS | 1 | 2
  CNS and PNS: Week 0: Abnormal, CS | 0 | 0
  CNS and PNS: Week 30: number analyzed (Participants) | 116 | 116
  CNS and PNS: Week 30: Normal | 115 | 115
  CNS and PNS: Week 30: Abnormal, NCS | 1 | 1
  CNS and PNS: Week 30: Abnormal, CS | 0 | 0
  CNS and PNS: Week 56: number analyzed (Participants) | 104 | 102
  CNS and PNS: Week 56: Normal | 104 | 101
  CNS and PNS: Week 56: Abnormal, NCS | 0 | 1
  CNS and PNS: Week 56: Abnormal, CS | 0 | 0
  CNS and PNS: Week 82: number analyzed (Participants) | 99 | 99
  CNS and PNS: Week 82: Normal | 99 | 98
  CNS and PNS: Week 82: Abnormal, NCS | 0 | 1
  CNS and PNS: Week 82: Abnormal, CS | 0 | 0
  Skin: Week 0: Normal | 76 | 58
  Skin: Week 0: Abnormal, NCS | 47 | 64
  Skin: Week 0: Abnormal, CS | 2 | 4
  Skin: Week 30: number analyzed (Participants) | 116 | 116
  Skin: Week 30: Normal | 71 | 56
  Skin: Week 30: Abnormal, NCS | 44 | 56
  Skin: Week 30: Abnormal, CS | 1 | 4
  Skin: Week 56: number analyzed (Participants) | 104 | 102
  Skin: Week 56: Normal | 65 | 48
  Skin: Week 56: Abnormal, NCS | 35 | 53
  Skin: Week 56: Abnormal, CS | 4 | 1
  Skin: Week 82: number analyzed (Participants) | 99 | 99
  Skin: Week 82: Normal | 57 | 50
  Skin: Week 82: Abnormal, NCS | 40 | 48
  Skin: Week 82: Abnormal, CS | 2 | 1
  Thyroid gland: Week 0: Normal | 124 | 124
  Thyroid gland: Week 0: Abnormal, NCS | 1 | 2
  Thyroid gland: Week 0: Abnormal, CS | 0 | 0
  Thyroid gland: Week 30: number analyzed (Participants) | 116 | 116
  Thyroid gland: Week 30: Normal | 115 | 114
  Thyroid gland: Week 30: Abnormal, NCS | 1 | 2
  Thyroid gland: Week 30: Abnormal, CS | 0 | 0
  Thyroid gland: Week 56: number analyzed (Participants) | 104 | 102
  Thyroid gland: Week 56: Normal | 103 | 101
  Thyroid gland: Week 56: Abnormal, NCS | 1 | 1
  Thyroid gland: Week 56: Abnormal, CS | 0 | 0
  Thyroid gland: Week 82: number analyzed (Participants) | 99 | 99
  Thyroid gland: Week 82: Normal | 97 | 98
  Thyroid gland: Week 82: Abnormal, NCS | 2 | 1
  Thyroid gland: Week 82: Abnormal, CS | 0 | 0
  Lymph node palpation: Week 0: Normal | 124 | 125
  Lymph node palpation: Week 0: Abnormal, NCS | 1 | 1
  Lymph node palpation: Week 0: Abnormal, CS | 0 | 0
  Lymph node palpation: Week 30: number analyzed (Participants) | 116 | 116
  Lymph node palpation: Week 30: Normal | 115 | 116
  Lymph node palpation: Week 30: Abnormal, NCS | 1 | 0
  Lymph node palpation: Week 30: Abnormal, CS | 0 | 0
  Lymph node palpation: Week 56: number analyzed (Participants) | 104 | 102
  Lymph node palpation: Week 56: Normal | 103 | 102
  Lymph node palpation: Week 56: Abnormal, NCS | 1 | 0
  Lymph node palpation: Week 56: Abnormal, CS | 0 | 0
  Lymph node palpation: Week 82: number analyzed (Participants) | 99 | 99
  Lymph node palpation: Week 82: Normal | 98 | 98
  Lymph node palpation: Week 82: Abnormal, NCS | 1 | 1
  Lymph node palpation: Week 82: Abnormal, CS | 0 | 0

59. Secondary Outcome: Change in Height SDS
Description: Change in height standard deviation score (SDS) was evaluated from baseline (week 0) to weeks 30 and 56, and from week 56 to week 82. Height SDS was calculated using the following formula: Z=[(value /M)^L - 1] / S*L; where L, M and S are median (M), skewness (L) and variation coefficient (S) of children/adolescents' height provided for each sex and age. For each subject, a standard deviation score Z (SDS) was calculated based on age and sex referring to the values L, M and S. The method is described in the WHO Multicentre Growth Reference, which also contains the values for L, M and S by age and sex. For Z (SDS) scores below -3 and above 3, the score was adjusted as described in the WHO instruction. Results are based on both participants who completed the trial period, week 0-30, week 0-56 or week 0-82, and participants who could not complete the corresponding trial period, but attended the follow-up visit at week 30, 56 or 82, respectively.
Time Frame: (Week 0, week 30); (Week 0, week 56); (Week 56, week 82)
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: SDS
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 125 | 126
SDS
  Change from week 0 to week 30: number analyzed (Participants) | 119 | 117
  Change from week 0 to week 30 | 0.11 (0.17) | 0.13 (0.18)
  Change from week 0 to week 56: number analyzed (Participants) | 115 | 105
  Change from week 0 to week 56 | 0.20 (0.27) | 0.24 (0.30)
  Change from week 56 to week 82: number analyzed (Participants) | 99 | 98
  Change from week 56 to week 82 | 0.07 (0.16) | 0.06 (0.12)

60. Secondary Outcome: Change in C-SSRS
Description: This outcome measure presents number of subjects with "suicidal ideation or suicidal behaviour on the Columbia Suicidality Severity Rating Scale (C-SSRS)" assessed at baseline (week 0), week 30, week 56 and week 82. Week 30, 56 and 82 results are based on the participants who completed the corresponding trial period, week 0-30, week 0-56 or week 0-82.
Time Frame: (Week 0, week 30); (Week 0, week 56); (Week 56, week 82)
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 125 | 126
Participants
  Wk 0: Suicidal ideation: number analyzed (Participants) | 122 | 126
  Wk 0: Suicidal ideation | 2 | 2
  Wk 0: Suicidal behaviour: number analyzed (Participants) | 122 | 126
  Wk 0: Suicidal behaviour | 0 | 1
  Wk0: Self-injurious behaviour, no suicidal intent: number analyzed (Participants) | 122 | 126
  Wk0: Self-injurious behaviour, no suicidal intent | 0 | 1
  Wk 30: Suicidal ideation: number analyzed (Participants) | 114 | 116
  Wk 30: Suicidal ideation | 0 | 0
  Wk 30: Suicidal behaviour: number analyzed (Participants) | 114 | 116
  Wk 30: Suicidal behaviour | 0 | 0
  Wk30: Self-injurious behaviour, no suicidal intent: number analyzed (Participants) | 114 | 116
  Wk30: Self-injurious behaviour, no suicidal intent | 0 | 0
  Wk 56: Suicidal ideation: number analyzed (Participants) | 101 | 100
  Wk 56: Suicidal ideation | 0 | 0
  Wk 56: Suicidal behaviour: number analyzed (Participants) | 101 | 100
  Wk 56: Suicidal behaviour | 0 | 0
  Wk56: Self-injurious behaviour, no suicidal intent: number analyzed (Participants) | 101 | 100
  Wk56: Self-injurious behaviour, no suicidal intent | 0 | 0
  Wk 82: Suicidal ideation: number analyzed (Participants) | 102 | 98
  Wk 82: Suicidal ideation | 0 | 0
  Wk 82: Suicidal behaviour: number analyzed (Participants) | 102 | 98
  Wk 82: Suicidal behaviour | 0 | 0
  Wk82: Self-injurious behaviour, no suicidal intent: number analyzed (Participants) | 102 | 97
  Wk82: Self-injurious behaviour, no suicidal intent | 0 | 0

61. Secondary Outcome: Change in PHQ-9
Description: Change in Patient Health Questionnaire 9 (PHQ-9) was evaluated from baseline (week 0) to weeks 30 and 56, and from week 56 to week 82. The PHQ-9 questionnaire is a 9-item depression module included in the patient health questionnaire, a self-administered diagnostic tool used for assessment of mental disorders. The PHQ-9 total score ranges from 0-27; total scores of 1-4 represent no depression, total scores of 5-9 represent mild depression, total scores of 10-14 represent moderate depression, total scores of 15-19 represent moderately severe depression and total scores of 20-27 represent severe depression. Results are based on the participants who completed the corresponding trial period, week 0-30, week 0-56 or week 0-82.
Time Frame: (Week 0, week 30); (Week 0, week 56); (Week 56, week 82)
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Liraglutide 3.0 mg | Placebo
Number analyzed (Participants) | 125 | 126
Score on a scale
  Change from week 0 to week 30: number analyzed (Participants) | 113 | 115
  Change from week 0 to week 30 | -1 (4) | -1 (4)
  Change from week 0 to week 56: number analyzed (Participants) | 102 | 100
  Change from week 0 to week 56 | -1 (3) | -2 (3)
  Change from week 56 to week 82: number analyzed (Participants) | 99 | 97
  Change from week 56 to week 82 | 0 (2) | -0 (3)

ADVERSE EVENTS:
Time Frame: Week 0-56 + 14 days. Results are based on the SAS which included all randomised participants exposed to at least one dose of trial product.
Description: All presented adverse events are TEAEs. A TEAE was defined as an event that occurred in the "on-treatment" period. 'On-treatment' period: Events with onset date between the first day of trial product administration and any of the following date, whichever came first: 1) 14 days after the last day on trial product, or 2) follow-up visit (week 58) for participants who discontinued trial product, or 3) last study visit (participants withdrawn without follow-up visit).
Arm/Group | Liraglutide 3.0 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 1/125 | 0/126
Serious Adverse Events (participants affected / at risk) | 3/125 | 5/126
Other Adverse Events (participants affected / at risk) | 100/125 | 84/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide 3.0 mg (N=125) | Placebo (N=126)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0)
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide 3.0 mg (N=125) | Placebo (N=126)
Abdominal pain (Gastrointestinal disorders) | 10 (15) | 11 (15)
Abdominal pain upper (Gastrointestinal disorders) | 17 (25) | 17 (23)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 8 (8)
Diarrhoea (Gastrointestinal disorders) | 28 (44) | 18 (29)
Dizziness (Nervous system disorders) | 13 (15) | 4 (5)
Dysmenorrhoea (Reproductive system and breast disorders) | 4 (5) | 8 (16)
Gastroenteritis (Infections and infestations) | 16 (22) | 6 (9)
Headache (Nervous system disorders) | 29 (43) | 35 (53)
Influenza (Infections and infestations) | 11 (11) | 12 (12)
Nasopharyngitis (Infections and infestations) | 34 (68) | 38 (80)
Nausea (Gastrointestinal disorders) | 53 (101) | 18 (25)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 15 (18)
Pharyngitis (Infections and infestations) | 4 (5) | 7 (7)
Pyrexia (General disorders) | 10 (11) | 9 (11)
Upper respiratory tract infection (Infections and infestations) | 11 (14) | 11 (16)
Vomiting (Gastrointestinal disorders) | 43 (85) | 5 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2019-12-11): https://cdn.clinicaltrials.gov/large-docs/79/NCT02918279/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-11): https://cdn.clinicaltrials.gov/large-docs/79/NCT02918279/SAP_001.pdf